CLINICAL TRIAL: NCT03207243
Title: A Randomized, Double-blind, Parallel Group, Multicenter, Stratified Study Evaluating the Efficacy and Safety of Repeat Doses of GSK3772847 Compared With Placebo in Participants With Moderately Severe Asthma
Brief Title: Efficacy and Safety Study of GSK3772847 in Subjects With Moderately Severe Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 207597; 2017-001072-34 (EudraCT Number)
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Results first posted 2020-03-02 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Asthma
Keywords: Severe asthma; Safety; GSK3772847; Efficacy
MeSH Terms: conditions — Asthma | interventions — melrilimab; Fluticasone-Salmeterol Drug Combination; Fluticasone

STUDY DESIGN:
Intervention Model Description: This will be a parallel intervention model in which GSK3772847 and placebo will be administered in parallel manner to randomized subjects.
Who Masked: Participant, Investigator
Masking Description: This is a double blind study and subjects and investigator will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Subjects receiving GSK3772847 (Experimental): Eligible subjects will receive GSK3772847 once every 4 weeks via IV route along with 500/50 mcg FP/Sal twice daily for first 2 weeks and dose of FP was reduced by approximately 50 percent at every 2 weeks until complete FP discontinuation.
  Interventions: Drug: GSK3772847; Drug: Fluticasone propionate/salmeterol; Drug: Fluticasone propionate
- Subjects receiving placebo drug (Placebo Comparator): Eligible subjects will receive placebo once every 4 weeks via IV route along with 500/50 mcg FP/Sal twice daily for first 2 weeks and dose of FP was reduced by approximately 50 percent at every 2 weeks until complete FP discontinuation.
  Interventions: Drug: Placebo; Drug: Fluticasone propionate/salmeterol; Drug: Fluticasone propionate

INTERVENTIONS:
Drug: GSK3772847 — GSK3772847 10 mg/kg will be administered as IV infusion once every 4 weeks to randomized subjects.
  Arms: Subjects receiving GSK3772847
Drug: Placebo — Placebo sterile normal saline will be administered as IV infusion once every 4 weeks to randomized subjects.
  Arms: Subjects receiving placebo drug
Drug: Fluticasone propionate/salmeterol — FP/Sal 500/50 mcg will be administered via inhalation route twice daily to all subjects.
Drug: Fluticasone propionate — FP 500, 250, 100 or 50 mcg will be administered via inhalation route twice daily to all subjects.

SUMMARY:
GSK3772847, an anti-interleukin (IL)33 receptor monoclonal antibody, is a novel treatment for asthma. This is a phase 2a study which aims to evaluate efficacy, safety, tolerability, pharmacokinetic (PK) and pharmacodynamic (PD) profiles of GSK3772847 in subjects with moderately severe asthma. The study will be conducted in 4 phases including screening, run-in phase, treatment phase and follow-up. In treatment phase, eligible subjects will be randomized to receive either GSK3772847 or placebo administered via intravenous (IV) route every 4 weeks in addition to open-label background therapy of fluticasone propionate/ salmeterol (FP/Sal) 500/50 micrograms (mcg) twice daily. During the treatment phase, the background therapy will be switched to FP 500 mcg for 2 weeks and the dose of FP will be reduced by approximately 50 percent at every 2 weeks until complete FP discontinuation. The total duration of study will be approximately 33 weeks and approximately 165 subjects with moderately severe asthma who are maintained on high-dose of inhaled corticosteroids/ Long-Acting Beta-2-Agonists (ICS/LABA) will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* Age: At least 18 years of age at the time of signing the informed consent.
* Males and females: A female subject is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: Not a woman of childbearing potential (WOCBP) OR A WOCBP who agrees to follow highly effective contraceptive methods from 4 weeks prior to the first dose of study medication and until at least 16 weeks after the last dose of study medication and completion of the follow-up visit.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.
* A subject with a documented diagnosis of moderate severe asthma based on Global Initiative for Asthma (GINA) 2016 Guidelines, whose asthma has been managed with regular treatment of high dose ICS defined as FP 500 mcg twice daily (i.e. 1000 mcg total daily dose) or equivalent, and LABA for at least 4 months. Additional therapy with a leukotriene receptor antagonist (LTRA) is permissible.
* Airway reversibility of at least 12 percent and 200 milliliter (mL) in FEV1 at Screening (Visit 1), or documented reversibility prior to Screening (Visit 1), or documented history of bronchial hyper reactivity (e.g. fall in FEV1 from baseline of more than or equal to 20percent with standard doses of methacholine or histamine, or more than or equal to 15 percent with standardized hyperventilation, hypertonic saline or mannitol challenge) from a bronchoprovocation study [e.g. methacholine challenge prior to Screening (Visit 1)].
* ACQ-5 score more than or equal to 1.0 and less than 4.0 at Screening (Visit 1).
* Had at least one asthma exacerbation within 12 months prior to screening that required treatment with systemic corticosteroid and/or hospitalization.
* All subjects must be able to replace their current Short-Acting Beta2-Agonists (SABA) treatment with albuterol/salbutamol aerosol inhaler at Visit 1 for use as needed, per product label, for the duration of the study.

Randomization inclusion criteria:

* ACQ-5 score more than or equal to 1.0 and less than 4.0 at Visit 2.
* Compliance with completion of the Daily eDiary reporting defined as completion of all questions/assessments on more than or equal to 4 of the last 7 days during the run-in period.

Exclusion Criteria:

* Current smokers or former smokers with a smoking history more than or equal to 10 pack years.
* Presence of a known pre-existing, clinically important respiratory conditions (e.g. pneumonia, pneumothorax, atelectasis segmental or larger, pulmonary fibrotic disease, bronchopulmonary dysplasia, chronic bronchitis, emphysema, chronic obstructive pulmonary disease, or other respiratory abnormalities) other than asthma.
* A pre-bronchodilator FEV1 less than 50 percent predicted of normal value at Screening (Visit 1).
* Subjects with a diagnosis of malignancy or in the process of investigation for a malignancy. Subjects with carcinoma that have not been in complete remission for at least 5 years. Subjects who have had carcinoma in situ of the cervix, squamous cell carcinoma and basal cell carcinoma of the skin would not be excluded based on the 5 year waiting period if the subject has been considered cured by treatment.
* Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at Screening (Visit 1) or within 3 months prior to first dose of study treatment.
* Site investigators will be provided with ECG over-read conducted by a centralized independent cardiologist, to assist in evaluation of subject eligibility.
* Weight: less than 50 kilograms (kg) and more than 150 kg.
* Regular use of systemic corticosteroids for conditions including asthma within 3 months prior to Screening (Visit 1).
* Subjects with high parasympathetic tone (e.g. trained athletes with baseline bradycardia) or chronic conditions associated with parasympathetic surges (e.g. migraines).
* Other conditions that could lead to elevated eosinophils such as hypereosinophilic syndromes. Subjects with a known, pre-existing parasitic infestation within 6 months prior to Screening (Visit 1).
* Clinically significant organic heart disease [e.g. Coronary artery disease (CAD), New York Heart Association (NYHA) Class III/IV heart failure].
* Ongoing infections (i.e. not resolved within 7 days prior to Screening [Visit 1]) or recurrent infections (i.e. requiring treatment for an identical diagnosis within 3 months) requiring systemic antibiotics Known, pre-existing parasitic infestations within 6 months prior to Screening.
* A subject must not have any clinically significant, uncontrolled condition, or disease state that, in the opinion of the investigator, would put the safety of the subject at risk through study participation or would confound the interpretation of the efficacy results if the condition/disease exacerbated during the study.
* A known immunodeficiency such as human immunodeficiency virus infection.
* Subjects with allergy or intolerance to a monoclonal antibody or biologic or to any components of the formulation used in this study.
* Subjects with a history (or suspected history) of alcohol misuse or substance abuse within 2 years prior to Screening (Visit 1).
* Subjects who are unable to follow study instructions such as visit schedule, dosing directions, study eDiary completion, or use of a standard metered dose inhaler. Subjects who have known evidence of lack of adherence to controller medication and/or ability to follow physician's recommendations. Any infirmity, disability, or geographic location that would limit compliance for scheduled visits.
* Subjects who have previously participated in a study of GSK3772847.
* Use of the prohibited medications is not permitted within the defined time intervals prior to Screening (Visit 1) and throughout the study. Potential subjects should not be washed out of their medication solely for the purpose on enrolling in the trial.
* A subject will not be eligible for this study if he/she is an immediate family member of the participating investigator, sub investigator, study coordinator, or employee of the participating investigator.
* In the opinion of the investigator, any subject who is unable to read and/or would not be able to complete a diary card/questionnaire.
* Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study.

Randomization exclusion criteria:

* Evidence of clinically significant abnormal laboratory tests during screening which are still abnormal upon repeat analysis and are not believed to be due to disease(s) present. Each Investigator will use his/her own discretion in determining the clinical significance of the abnormality.
* Evidence of clinically significant abnormal ECG findings at Visit 2.
* An abnormal and significant finding from 24-hour Holter monitoring at Screening (Visit 1). Investigators will be provided with Holter reviews conducted by an independent cardiologist to assist in evaluation of subject eligibility.
* Liver function at screening (Visit 1): ALT more than 2 x upper limit of normal (ULN) and bilirubin more than 1.5xULN (isolated bilirubin more than 1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin less than 35 percent); Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Subjects with ongoing asthma exacerbation at the time of Visit 2.
* A pre-bronchodilator FEV1 less than 50 percent predicted of normal value at Visit 2.
* Positive pregnancy test at Visit 0, Screening (Visit 1) or Visit 2.
* Ongoing or recurrent infections requiring systemic antibiotics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (52):
- United States (27):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Scottsboro, Alabama
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Winter Park, Florida
  - GSK Investigational Site, Adairsville, Georgia
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Mooresville, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Boerne, Texas
  - GSK Investigational Site, Williamsburg, Virginia
  - GSK Investigational Site, Madison, Wisconsin
- Australia (4):
  - GSK Investigational Site, Woodville South, South Australia
  - GSK Investigational Site, Clayton, Victoria
  - GSK Investigational Site, Melbourne, Victoria
  - GSK Investigational Site, Parkville, Victoria
- Canada (7):
  - GSK Investigational Site, Sherwood Park, Alberta
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Trois-Rivières, Quebec
  - GSK Investigational Site, Québec
- Mexico (7):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Cuernavaca, Morelos
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, Villahermosa, Tabasco
  - GSK Investigational Site, Mérida, Yucatán
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, México DF
- Russia (6):
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Samara
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Ulyanovsk
- GSK Investigational Site, Kyiv, Ukraine

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, double-blind, placebo-controlled, parallel-group multicenter study to assess the efficacy, safety and tolerability, pharmacokinetic (PK) and pharmacodynamic (PD) profiles of GSK3772847 in participants with moderately severe asthma.
Pre-assignment Details: A total of 165 participants with moderately severe asthma were randomized to receive GSK3772847 or placebo.
Groups:
- Placebo: Participants were administered placebo via intravenous (IV) route every 4 weeks (Weeks 0, 4, 8 and 12) in addition to open-label background therapy of fluticasone propionate/ salmeterol (FP/Sal) 500/50 micrograms (mcg) twice daily. After 2 weeks, the background therapy was switched to FP 500 mcg for 2 weeks and the dose of FP was reduced by approximately 50 percent at every 2 weeks until complete FP discontinuation. Three Follow-up visits were performed after the End of Treatment Period (ETP) Visit (Weeks 20, 24, and 28) for safety assessments. Participants received salbutamol/albuterol to use as needed for asthma symptom relief.
- GSK3772847: Participants were administered 10 milligram/kilogram (mg/kg) GSK3772847 via IV route every 4 weeks (Weeks 0, 4, 8 and 12) in addition to open-label background therapy of FP/Sal 500/50 mcg twice daily. After 2 weeks, the background therapy was switched to FP 500 mcg for 2 weeks and the dose of FP was reduced by approximately 50 percent at every 2 weeks until complete FP discontinuation. Three Follow-up visits were performed after the ETP Visit (Weeks 20, 24, and 28) for safety assessments. Participants received salbutamol/albuterol to use as needed for asthma symptom relief.
Period: Overall Study
Arm/Group | Placebo | GSK3772847
Started | 82 | 83
Completed | 23 | 39
Not Completed | 59 | 44
Not completed — Adverse Event | 2 | 2
Not completed — Loss of Asthma Control | 47 | 31
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Physician Decision | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Specified Withdrawal Criteria | 7 | 2
Not completed — Protocol Violation | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK3772847 | Total
Number analyzed (Participants) | 82 | 83 | 165
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.1 (11.65) | 51.8 (11.74) | 52.9 (11.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 64 | 118
  Male | 28 | 19 | 47
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 14 | 8 | 22
  Central/South Asian Heritage | 0 | 1 | 1
  Japanese /East Asian/South East Asian Heritage | 1 | 0 | 1
  Black or African American | 3 | 8 | 11
  White | 64 | 66 | 130

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Loss of Asthma Control Over Weeks 0-16
Description: Loss of asthma control is defined as: Asthma Control Questionnaire (ACQ-5) score increase from Baseline >=0.5 point or pre-bronchodilator forced expiratory volume in 1 second (FEV1) decrease from baseline >7.5 % or inability to titrate inhaled corticosteroid or a clinically significant asthma exacerbation (requiring oral corticosteroid [OCS] and/or hospitalization). The analysis shown is for primary estimand which includes all data collected, except for data collected after the date of loss of asthma control or early withdrawal from study treatment. Baseline is defined as Day1. Percentage of participants experiencing loss of asthma control up to Week 16 has been presented. Modified Intent-to-Treat (Loss of Control) (mITT_LoC) population consisted of all randomized participants who took at least 1 dose of study treatment and if participants experienced loss of asthma control, they were analyzed according to actual treatment at time of loss of control.
Time Frame: Up to Week 16
Population: Modified Intent-to-Treat (Loss of Control) (mITT_LoC) Population. Only those participants with data available at indicated time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 70 | 70
Percentage of participants | 81 | 67
Statistical Analysis 1: Comparison: Placebo vs GSK3772847; Test type: Other; Median Rate Ratio = 0.82, 95% CI 2-sided [0.66 to 0.99] — Median rate ratio (Placebo - GSK3772847) and its 95% Credible Interval has been presented

2. Secondary Outcome: Percentage of Participants With >=0.5 Point Asthma Control Questionnaire (ACQ-5) Score Increase From Baseline
Description: The ACQ-5 is a five-item, self-completed questionnaire, which measures asthma control of a participant. The five questions (concerning nocturnal awakening, waking in the morning, activity limitation, shortness of breath and wheeze) enquire about the frequency and/or severity of symptoms over the previous week. The response options for all these questions range from zero (no impairment/limitation) to six (total impairment/ limitation) scale. ACQ-5 score ranges from 0 (totally controlled) to 6 (severely uncontrolled). Higher score indicate lower asthma control. Baseline is the latest available assessment prior to first dose (Day 1). Change from Baseline was calculated by subtracting Baseline value from the specified time point value. A change of >=0.5 in score suggests a clinically important change in score. Data is presented for primary estimand which includes all data collected, except for data collected after the date of loss of asthma control or early withdrawal from study treatment
Time Frame: Baseline and up to Week 16
Population: Modified Intent-to-Treat (Loss of Control) Population. Only those participants with data available at indicated time points who experienced loss of asthma control were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 57 | 47
Percentage of participants | 39 | 30

3. Secondary Outcome: Percentage of Participants Who Have Pre-bronchodilator FEV1 Decrease From Baseline >7.5 %
Description: Pulmonary function is measured by FEV1. FEV1 is the amount of air expired in 1 second. Pre-bronchodilator FEV1 measurements were taken by spirometry. Baseline is defined as the latest available pre-dose assessment (Day 1). Decrease from Baseline >7.5 % in score suggests worsening of condition.
Time Frame: Baseline and up to Week 16
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 57 | 47
Percentage of participants | 63 | 68

4. Secondary Outcome: Percentage of Participants With Inability to Titrate Inhaled Corticosteroids (ICS)
Description: Corticosteroid titration allows overall clinical evaluation of the participant's asthma status taking into account both lung function and symptom control. Inability to titrate inhaled corticosteroids indicates loss of asthma control.
Time Frame: Up to Week 16
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 57 | 47
Percentage of participants | 23 | 30

5. Secondary Outcome: Percentage of Participants With Clinically Significant Asthma Exacerbation
Description: A clinically significant asthma exacerbation is defined as one requiring oral corticosteroid and/or hospitalization.
Time Frame: Up to Week 16
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 57 | 47
Percentage of participants | 7 | 13

6. Secondary Outcome: Percentage of Participants With Loss of Asthma Control Over Weeks 0-6
Description: Loss of asthma control is defined as: ACQ-5 score increase from Baseline >=0.5 point or pre-bronchodilator FEV1 decrease from Baseline >7.5 % or inability to titrate inhaled corticosteroid or a clinically significant asthma exacerbation (requiring oral OCS and/or hospitalization). The analysis shown is for primary estimand which includes all data collected, except for data collected after the date of loss of asthma control or early withdrawal from study treatment. Baseline is defined as Day1. Percentage of participants experiencing loss of asthma control up to Week 6 has been presented.
Time Frame: Up to Week 6
Population: Modified Intent-to-Treat (Loss of Control) Population. Only those participants with data available at indicated time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 70 | 72
Percentage of participants | 50 | 36
Statistical Analysis 1: Comparison: Placebo vs GSK3772847; Test type: Other; Median Rate Ratio = 0.71, 95% CI 2-sided [0.44 to 1.01] — Median rate ratio (Placebo - GSK3772847) and its 95% Credible Interval has been presented

7. Secondary Outcome: Time to Loss of Asthma Control
Description: Time to loss of asthma control was analyzed using Kaplan-Meier analysis. In this analysis, participants were either be counted as an event or they were censored. An event is defined as participants who experience loss of asthma control during the study. Censoring is defined as participants who discontinued investigational product for reasons other than loss of asthma control. The analysis shown is for primary estimand which includes all data collected, except for data collected after the date of loss of asthma control or early withdrawal from study treatment. Participants who didn't experience loss of asthma control were also censored at day 113.
Time Frame: Up to Week 16
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 57 | 47
Days | 50 [29 to NA] — NA indicates data could not be calculated due to insufficient number of participants with events. | 96 [31 to NA] — NA indicates data could not be calculated due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Placebo vs GSK3772847; Test type: Other; p = 0.044, Log Rank

8. Secondary Outcome: Percentage of Participants With Clinically Significant Asthma Exacerbation or Inability to Titrate
Description: A clinically significant asthma exacerbation is defined as one requiring oral corticosteroid and/or hospitalization. Participants with clinically significant asthma exacerbation or inability to titrate FP indicated loss of asthma control.
Time Frame: Up to Week 16
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 57 | 47
Percentage of participants | 25 | 40

9. Secondary Outcome: Number of Participants Experiencing Asthma Related Hospitalization During the Study Period
Description: Hospitalization is defined as an inpatient stay or least an overnight stay at the hospital or emergency ward for observation or other equivalent facility. Data has been presented for primary estimand which includes all data collected, except for data collected after the date of loss of asthma control or early withdrawal from study treatment.
Time Frame: Up to Week 16
Population: Modified Intent-to-Treat (mITT) population consisted of all randomized participants who took at least 1 dose of study treatment and were analyzed according to the treatment they received >=50% of the time.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 78 | 78
Participants | 1 | 0

10. Secondary Outcome: Rate Per 1000 Person-years of Participants With Hospitalization
Description: An event is defined as an on-treatment asthma-related hospitalization or emergency room visit and participants can contribute to more than one event. Rate is calculated as number of events * 1000 divided by (number of participants in treatment group * mean treatment exposure in years). Data has been presented for primary estimand which includes all data collected, except for data collected after the date of loss of asthma control or early withdrawal from study treatment.
Time Frame: Up to Week 16
Population: Modified Intent-to-Treat Population.
Measure: Number; unit: Events per person-year
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 78 | 78
Events per person-year | 70.5 | 0

11. Secondary Outcome: Number of Hospitalizations or Emergency Room Visits Per Participants
Description: The number of hospitalization or emergency room visit made by per participant due to loss of asthma control have been presented in category titles. Data has been presented for primary estimand which includes all data collected, except for data collected after the date of loss of asthma control or early withdrawal from study treatment.
Time Frame: Up to Week 16
Population: Modified Intent-to-Treat Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 78 | 78
Participants
  0 | 77 | 78
  1 | 1 | 0
  2 | 0 | 0
  >=3 | 0 | 0

12. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire (ACQ-5) Total Score
Description: ACQ-5 is a five-item, self-completed questionnaire, which measures asthma control of a participant. The five questions (concerning nocturnal awakening, waking in the morning, activity limitation, shortness of breath & wheeze) enquire about the frequency &/or severity of symptoms over the previous week. The response options range from zero (no impairment/limitation) to six (total impairment/limitation) scale. ACQ-5 score ranges from 0 (totally controlled) to 6 (severely uncontrolled). Higher score indicate lower asthma control. Baseline is the latest available assessment prior to first dose (Day 1). Change from Baseline was calculated by subtracting Baseline value from the specified time point value. Data is presented for primary estimand which includes all data collected, except for data collected after the date of loss of asthma control or early withdrawal from study treatment.
Time Frame: Baseline and Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15 and Week 16
Population: Modified Intent-to-Treat Population. Only those participants with data available at indicated time points were analyzed. Participants with data available at specified time points were represented by n=x in the category titles.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 72 | 73
Scores on a scale
  Week1; n=72, 73 | -0.36 (0.713) | -0.48 (0.685)
  Week2; n=67, 68: number analyzed (Participants) | 67 | 68
  Week2; n=67, 68 | -0.53 (0.666) | -0.74 (0.732)
  Week3; n=61, 61: number analyzed (Participants) | 61 | 61
  Week3; n=61, 61 | -0.59 (0.722) | -0.78 (0.663)
  Week4; n=54, 59: number analyzed (Participants) | 54 | 59
  Week4; n=54, 59 | -0.69 (0.733) | -0.79 (0.695)
  Week5; n= 42, 52: number analyzed (Participants) | 42 | 52
  Week5; n= 42, 52 | -0.80 (0.839) | -0.78 (0.804)
  Week6; n=40, 48: number analyzed (Participants) | 40 | 48
  Week6; n=40, 48 | -0.80 (0.907) | -0.93 (0.692)
  Week7; n=34, 46: number analyzed (Participants) | 34 | 46
  Week7; n=34, 46 | -0.92 (0.710) | -0.93 (0.785)
  Week8; n=33, 44: number analyzed (Participants) | 33 | 44
  Week8; n=33, 44 | -0.95 (0.769) | -1.00 (0.755)
  Week9; n=30, 42: number analyzed (Participants) | 30 | 42
  Week9; n=30, 42 | -0.93 (0.713) | -0.97 (0.817)
  Week10; n=29, 41: number analyzed (Participants) | 29 | 41
  Week10; n=29, 41 | -0.97 (0.820) | -0.99 (0.729)
  Week11; n=22, 38: number analyzed (Participants) | 22 | 38
  Week11; n=22, 38 | -1.05 (0.907) | -1.07 (0.770)
  Week12; n=23, 38: number analyzed (Participants) | 23 | 38
  Week12; n=23, 38 | -0.88 (1.134) | -1.16 (0.795)
  Week13; n=17,32: number analyzed (Participants) | 17 | 32
  Week13; n=17,32 | -1.40 (0.860) | -1.06 (0.773)
  Week14; n=17, 31: number analyzed (Participants) | 17 | 31
  Week14; n=17, 31 | -1.33 (0.943) | -1.14 (0.820)
  Week15; n=17, 27: number analyzed (Participants) | 17 | 27
  Week15; n=17, 27 | -1.22 (0.874) | -1.21 (0.814)
  Week16; n=12, 21: number analyzed (Participants) | 12 | 21
  Week16; n=12, 21 | -1.15 (1.102) | -1.17 (0.738)

13. Secondary Outcome: Percentage of Participants With <=-0.5 Point ACQ-5 Score Decrease From Baseline (Responder)
Description: ACQ-5 is a five-item, self-completed questionnaire, which measures asthma control of a participant. The five questions (concerning nocturnal awakening, waking in the morning, activity limitation, shortness of breath & wheeze) enquire about the frequency &/or severity of symptoms over the previous week. The response options range from zero (no impairment/limitation) to six (total impairment/limitation) scale. ACQ-5 score ranges from 0 (totally controlled) to 6 (severely uncontrolled). Higher score indicate lower asthma control. Baseline is the latest available assessment prior to first dose (Day 1). Change from Baseline was calculated by subtracting Baseline value from the specified time point value. A responder is defined as participants with change from Baseline of <= -0.5 point at given time point. Data is presented for primary estimand which includes all data collected, except for data collected after the date of loss of asthma control or early withdrawal from study treatment.
Time Frame: Baseline and Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15 and Week 16
Population: as for outcome 12
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 72 | 73
Percentage of participants
  Week1; n=72, 73 | 38 | 41
  Week2; n=67, 68: number analyzed (Participants) | 67 | 68
  Week2; n=67, 68 | 46 | 56
  Week3; n=61, 61: number analyzed (Participants) | 61 | 61
  Week3; n=61, 61 | 49 | 56
  Week4; n=54, 59: number analyzed (Participants) | 54 | 59
  Week4; n=54, 59 | 59 | 61
  Week5; n= 42, 52: number analyzed (Participants) | 42 | 52
  Week5; n= 42, 52 | 62 | 65
  Week6; n=40, 48: number analyzed (Participants) | 40 | 48
  Week6; n=40, 48 | 63 | 69
  Week7; n=34, 46: number analyzed (Participants) | 34 | 46
  Week7; n=34, 46 | 74 | 65
  Week8; n=33, 44: number analyzed (Participants) | 33 | 44
  Week8; n=33, 44 | 70 | 73
  Week9; n=30, 42: number analyzed (Participants) | 30 | 42
  Week9; n=30, 42 | 70 | 71
  Week10; n=29, 41: number analyzed (Participants) | 29 | 41
  Week10; n=29, 41 | 69 | 76
  Week11; n=22, 38: number analyzed (Participants) | 22 | 38
  Week11; n=22, 38 | 64 | 79
  Week12; n=23, 38: number analyzed (Participants) | 23 | 38
  Week12; n=23, 38 | 57 | 79
  Week13; n=17,32: number analyzed (Participants) | 17 | 32
  Week13; n=17,32 | 82 | 75
  Week14; n=17, 31: number analyzed (Participants) | 17 | 31
  Week14; n=17, 31 | 71 | 74
  Week15; n=17, 27: number analyzed (Participants) | 17 | 27
  Week15; n=17, 27 | 76 | 74
  Week16; n=12, 21: number analyzed (Participants) | 12 | 21
  Week16; n=12, 21 | 67 | 81

14. Secondary Outcome: Change From Baseline in St George's Respiratory Questionnaire (SGRQ) Total Score
Description: SGRQ is a disease-specific questionnaire designed to measure impact of respiratory disease and its treatment on Health-related quality of life (HRQoL) of participants with Chronic Obstructive Pulmonary Disease (COPD). It contains 14 questions with a total of 40 items grouped into domains (Symptoms, Activity and Impacts). SGRQ total score was calculated as 100 multiplied by summed weights from all positive items divided by sum of weights for all items in questionnaire. It ranges from 0 to 100, higher score indicates poor HRQoL. Baseline is defined as the latest available assessment prior to first dose (Day 1). Change from Baseline was calculated by subtracting Baseline value from the specified time point value. Data is presented for primary estimand which includes all data collected, except for data collected after the date of loss of asthma control or early withdrawal from study treatment.
Time Frame: Baseline and Weeks 4, 8, 12 and 16
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 43 | 52
Scores on a scale
  Week4; n=43, 52 | -10.0 (14.98) | -7.0 (11.41)
  Week8; n=31, 42: number analyzed (Participants) | 31 | 42
  Week8; n=31, 42 | -10.7 (15.32) | -7.2 (17.08)
  Week12; n=23, 35: number analyzed (Participants) | 23 | 35
  Week12; n=23, 35 | -15.8 (21.42) | -12.9 (14.91)
  Week16; n=16, 26: number analyzed (Participants) | 16 | 26
  Week16; n=16, 26 | -12.4 (20.75) | -16.5 (18.51)

15. Secondary Outcome: Percentage of Participants With at Least a 4 Units Improvement From Baseline of St. George's Respiratory Questionnaire (SGRQ)
Description: SGRQ is a disease-specific questionnaire designed to measure impact of respiratory disease and its treatment on HRQoL of participants with COPD. It contains 14 questions with a total of 40 items grouped into domains (Symptoms, Activity and Impacts). SGRQ total score was calculated as 100 multiplied by summed weights from all positive items divided by sum of weights for all items in questionnaire. It ranges from 0 to 100, higher score indicates poor HRQoL. Baseline is defined as the latest available assessment prior to first dose (Day 1). A responder is defined as a change from Baseline of <= -4 at the given time point. Data is presented for primary estimand which includes all data collected, except for data collected after the date of loss of asthma control or early withdrawal from study treatment.
Time Frame: Baseline and Weeks 4, 8, 12 and 16
Population: Modified Intent-to-Treat Population. Only those participants with data available at the indicated time points were analyzed. Participants with data available at specified time points were represented by n=x in the category titles.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 43 | 52
Percentage of participants
  Week4; n=43, 52 | 60 | 58
  Week8; n=31, 42: number analyzed (Participants) | 31 | 42
  Week8; n=31, 42 | 61 | 67
  Week12; n=23, 35: number analyzed (Participants) | 23 | 35
  Week12; n=23, 35 | 70 | 74
  Week16; n=16, 26: number analyzed (Participants) | 16 | 26
  Week16; n=16, 26 | 69 | 88

16. Secondary Outcome: Change From Baseline in Pre-bronchodilator Forced Expiratory Volume in One Second (FEV1)
Description: Pre-bronchodilator FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Baseline is defined as the latest available assessment prior to first dose (Day 1) and change from Baseline was calculated by subtracting Baseline value from the specified time point value. Data is presented for primary estimand which includes all data collected, except for data collected after the date of loss of asthma control or early withdrawal from study treatment.
Time Frame: Baseline and Weeks 2, 4, 6, 8, 10, 12, 14 and 16
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 64 | 66
Liters
  Week2; n=64, 66 | 0.094 (0.2359) | 0.089 (0.2443)
  Week4; n=48, 56: number analyzed (Participants) | 48 | 56
  Week4; n=48, 56 | 0.074 (0.3077) | 0.086 (0.2325)
  Week6; n=38, 50: number analyzed (Participants) | 38 | 50
  Week6; n=38, 50 | 0.078 (0.2610) | 0.135 (0.3758)
  Week8; n=33, 45: number analyzed (Participants) | 33 | 45
  Week8; n=33, 45 | 0.049 (0.2888) | 0.089 (0.2236)
  Week10; n=33, 43: number analyzed (Participants) | 33 | 43
  Week10; n=33, 43 | 0.047 (0.2563) | 0.066 (0.2372)
  Week12; n=23, 36: number analyzed (Participants) | 23 | 36
  Week12; n=23, 36 | 0.061 (0.2759) | 0.037 (0.2637)
  Week14; n=21, 36: number analyzed (Participants) | 21 | 36
  Week14; n=21, 36 | 0.079 (0.2824) | 0.047 (0.3200)
  Week16; n=15, 26: number analyzed (Participants) | 15 | 26
  Week16; n=15, 26 | 0.063 (0.3383) | 0.025 (0.3008)

17. Secondary Outcome: Change From Baseline in Mean Morning Peak Expiratory Flow (PEF) and Mean Evening PEF
Description: PEF is maximum speed of expiration measured, using spirometer. The device was distributed to participants at Visit 1, to measure PEF twice-daily (morning upon waking & in the evening just before going to bed). Participants were encouraged to perform morning & evening PEF measurements before the use of any long-acting beta-agonists (LABAs) or rescue medication. Highest of 3 values were recorded in eDairy.Baseline was calculated over the last 7 days of run-in period prior to Visit 2 (Week 0). Participants with at least 4 full days of data in the last 7 days of run-in were included. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. Mean PEF was calculated for each participant during the four weekly periods (Weeks 1-4; Weeks 5-8, Weeks 9-12 and Weeks 13-16).Data is presented for primary estimand which includes all data collected, except for data collected after the date of loss of asthma control or early withdrawal from study treatment
Time Frame: Baseline and Weeks 1-4; Weeks 5-8, Weeks 9-12 and Weeks 13-16.
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Liters/minute
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 76 | 77
Liters/minute
  Morning PEF: Weeks 1-4,n=76, 76: number analyzed (Participants) | 76 | 76
  Morning PEF: Weeks 1-4,n=76, 76 | 4.13 (35.492) | 4.32 (43.773)
  Morning PEF: Weeks 5-8,n=50, 56: number analyzed (Participants) | 50 | 56
  Morning PEF: Weeks 5-8,n=50, 56 | -1.84 (65.222) | -3.82 (46.621)
  Morning PEF: Weeks 9-12,n=31, 43: number analyzed (Participants) | 31 | 43
  Morning PEF: Weeks 9-12,n=31, 43 | -4.15 (46.588) | -1.69 (45.192)
  Morning PEF: Weeks 13-16,n=20, 38: number analyzed (Participants) | 20 | 38
  Morning PEF: Weeks 13-16,n=20, 38 | -7.88 (47.190) | -1.83 (69.866)
  Evening PEF: Weeks 1-4,n=76, 77 | 0.43 (36.087) | 2.45 (37.712)
  Evening PEF: Weeks 5-8,n=52, 58: number analyzed (Participants) | 52 | 58
  Evening PEF: Weeks 5-8,n=52, 58 | -6.96 (61.987) | -4.38 (49.076)
  Evening PEF: Weeks 9-12,n=33, 44: number analyzed (Participants) | 33 | 44
  Evening PEF: Weeks 9-12,n=33, 44 | -0.77 (54.768) | -0.58 (39.929)
  Evening PEF: Weeks 13-16,n=21, 38: number analyzed (Participants) | 21 | 38
  Evening PEF: Weeks 13-16,n=21, 38 | -10.81 (51.566) | -1.16 (63.383)

18. Secondary Outcome: Change From Baseline in Mean Daytime Asthma Symptom Score Over Each Four Weeks of the 16 Week Treatment Period
Description: Asthma symptoms experienced by participants during the day was recorded in e-Diary every evening before going to bed in form of scores on a 5-point rating scale. Scores ranged from 0=no daytime asthma symptoms to 4=very severe daytime asthma symptoms. Baseline was calculated over the last 7 days of run-in period prior to Visit 2 (Week 0). Participants with at least 4 full days of data in the last 7 days of run-in were included. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. The mean asthma symptom score was calculated for each participant during the four weekly periods (Weeks 1-4; Weeks 5-8, Weeks 9-12 and Weeks 13-16). Data is presented for primary estimand which includes all data collected, except for data collected after the date of loss of asthma control or early withdrawal from study treatment.
Time Frame: Baseline and Weeks 1-4; Weeks 5-8, Weeks 9-12 and Weeks 13-16
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 77 | 78
Scores on a scale
  Weeks 1-4, n=77, 78 | -0.09 (0.472) | -0.02 (0.337)
  Weeks 5-8, n=52, 59: number analyzed (Participants) | 52 | 59
  Weeks 5-8, n=52, 59 | -0.18 (0.610) | -0.09 (0.460)
  Weeks 9-12 ,n=33,34: number analyzed (Participants) | 33 | 34
  Weeks 9-12 ,n=33,34 | -0.29 (0.631) | -0.08 (0.473)
  Weeks 13-16, n=21, 38: number analyzed (Participants) | 21 | 38
  Weeks 13-16, n=21, 38 | -0.29 (0.692) | -0.17 (0.458)

19. Secondary Outcome: Change From Baseline in Mean Daily Rescue Medication Use (Albuterol/Salbutamol)
Description: The mean number of inhalation of rescue medication (albuterol/salbutamol) used to relieve symptoms immediately during the day and night was recorded in eDiary from Baseline until Week 16. Baseline was calculated over the last 7 days of run-in period prior to Visit 2 (Week 0). Participants with at least 4 full days of data in the last 7 days of run-in were included. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. The mean rescue medication use was calculated for each participant during the four weekly periods (Weeks 1-4; Weeks 5-8, Weeks 9-12 and Weeks 13-16). Data is presented for primary estimand which includes all data collected, except for data collected after the date of loss of asthma control or early withdrawal from study treatment.
Time Frame: Baseline and Weeks 1-4; Weeks 5-8, Weeks 9-12 and Weeks 13-16
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Inhalations per day
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 78 | 75
Inhalations per day
  Weeks 1-4, n=78, 75 | -0.52 (2.554) | -1.09 (4.687)
  Weeks 5-8, n=56, 57: number analyzed (Participants) | 56 | 57
  Weeks 5-8, n=56, 57 | -0.52 (1.740) | -1.24 (5.180)
  Weeks 9-12, n=32, 42: number analyzed (Participants) | 32 | 42
  Weeks 9-12, n=32, 42 | -0.17 (0.945) | -1.59 (5.934)
  Weeks 13-16, n=24, 37: number analyzed (Participants) | 24 | 37
  Weeks 13-16, n=24, 37 | 0.01 (2.005) | -1.90 (6.624)

20. Secondary Outcome: Change From Baseline in Percent Night-time Awakenings Due to Asthma Symptoms Requiring Rescue Medication Use
Description: Participant captured night-time awakenings (yes/no) and use of rescue medication during these awakenings (yes/no) was recorded in e-Diary each morning. Percentage of night-time awakenings is calculated by number of nights with awakenings due to asthma and requiring rescue medication divided by number of nights with data available*100. Baseline was calculated over the last 7 days of run-in period prior to Visit 2 (Week 0). Participants having at least 4 full days of data in the last 7 days of run-in were included. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. Night-time awakenings due to asthma symptoms requiring rescue medication was calculated for each participant during the four weekly periods (Weeks 1-4; Weeks 5-8, Weeks 9-12 and Weeks 13-16). Data is presented for primary estimand which includes all data collected, except for data collected after the date of loss of asthma control or early withdrawal from study treatment.
Time Frame: Baseline and Weeks 1-4; Weeks 5-8, Weeks 9-12 and Weeks 13-16
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Percentage of nights with awakenings
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 77 | 76
Percentage of nights with awakenings
  Weeks 1-4, n=77, 76 | -3.80 (25.712) | -7.42 (23.847)
  Weeks 5-8,n=50, 56: number analyzed (Participants) | 50 | 56
  Weeks 5-8,n=50, 56 | -7.85 (26.325) | -10.49 (31.081)
  Weeks 9-12,n=31, 43: number analyzed (Participants) | 31 | 43
  Weeks 9-12,n=31, 43 | -5.67 (24.669) | -13.43 (26.962)
  Weeks 13-16,n=20, 38: number analyzed (Participants) | 20 | 38
  Weeks 13-16,n=20, 38 | -2.31 (30.355) | -14.91 (33.544)

21. Secondary Outcome: Percent Change From Baseline in Fractional Exhaled Nitric Oxide (FeNO)
Description: FeNO was assessed as a measure of airway inflammation using a handheld electronic device. The measurements recorded were according to standardized procedures by the American Thoracic Society and the European Respiratory Society Recommendations for Standardized Procedures for the Online and Offline Measurement of Exhaled Lower Respiratory Nitric Oxide and Nasal Nitric Oxide. FeNO measurements were obtained prior to FEV1 assessments. Participants did not use their rescue medication for at least 6 hours before each FeNO assessment, unless essential for clinical need. Baseline is defined as the latest available assessment prior to first dose (Day 1). Percent change from Baseline is calculated as ratio to Baseline minus one and multiplied by 100. Data is presented for primary estimand which includes all data collected, except for data collected after the date of loss of asthma control or early withdrawal from study treatment.
Time Frame: Baseline and Weeks 1, 2, 4, 6, 8, 10, 12, 14 and 16
Population: as for outcome 12
Measure: Median (Full Range); unit: Percent Change
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 60 | 63
Percent Change
  Week1; n=60, 63 | -3.6 [-46 to 126] | -4.9 [-57 to 281]
  Week2; n=58, 59: number analyzed (Participants) | 58 | 59
  Week2; n=58, 59 | 15.4 [-57 to 481] | 0.0 [-66 to 206]
  Week4; n=41, 50: number analyzed (Participants) | 41 | 50
  Week4; n=41, 50 | 15.2 [-64 to 302] | 3.3 [-69 to 546]
  Week6; n=34, 46: number analyzed (Participants) | 34 | 46
  Week6; n=34, 46 | 5.0 [-71 to 537] | 0.0 [-62 to 221]
  Week8; n=29, 38: number analyzed (Participants) | 29 | 38
  Week8; n=29, 38 | 15.9 [-60 to 548] | -2.9 [-40 to 148]
  Week10; n=29, 37: number analyzed (Participants) | 29 | 37
  Week10; n=29, 37 | 13.8 [-54 to 483] | 0.0 [-52 to 252]
  Week12; n=19, 31: number analyzed (Participants) | 19 | 31
  Week12; n=19, 31 | 31.4 [-40 to 422] | 8.8 [-47 to 413]
  Week14; n=19, 30: number analyzed (Participants) | 19 | 30
  Week14; n=19, 30 | 28.1 [-43 to 483] | 1.7 [-48 to 457]
  Week16; n=13, 22: number analyzed (Participants) | 13 | 22
  Week16; n=13, 22 | 85.9 [-33 to 635] | 12.7 [-51 to 695]

22. Secondary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs) and Non-Serious Adverse Events (Non-SAEs)
Description: A non-SAE is any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment were categorized as SAE.
Time Frame: Up to Week 16
Population: Safety Population consists of all randomized participants who took at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 82 | 83
Participants
  non-SAE | 20 | 19
  SAE | 1 | 2

23. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)
Description: DBP and SBP were measured in semi-supine position after 5 minutes rest. Baseline is defined as the most recent recorded value before dosing on Day 1. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. Data for change from Baseline for post dose values have been presented.
Time Frame: Baseline and Week 0 (Post-dose), Week1, Week 2, Week 4 (Pre and Post dose), Week 6, Week 8 (Pre and Post dose), Week 10, Week 12 (Pre and Post dose), Week 14, Week 16, Week 20, Week 24 and Week 28
Population: Safety Population. Participants with data available at specified time points were represented by n=x in the category titles.
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 82 | 83
Millimeters of Mercury (mmHg)
  SBP: Post-dose: Week0; n=82, 83 | -2.0 (8.05) | 1.3 (7.19)
  SBP: Week1; n=79, 75: number analyzed (Participants) | 79 | 75
  SBP: Week1; n=79, 75 | -0.9 (9.61) | 0.4 (9.67)
  SBP: Week2; n=73, 75: number analyzed (Participants) | 73 | 75
  SBP: Week2; n=73, 75 | -1.3 (10.73) | -1.3 (10.58)
  SBP: Pre-dose: Week4; n=49, 59: number analyzed (Participants) | 49 | 59
  SBP: Pre-dose: Week4; n=49, 59 | -2.0 (8.88) | -0.1 (8.84)
  SBP: Post-dose: Week4; n=48, 59: number analyzed (Participants) | 48 | 59
  SBP: Post-dose: Week4; n=48, 59 | -2.0 (9.46) | 2.2 (10.72)
  SBP:Week6; n=45, 57: number analyzed (Participants) | 45 | 57
  SBP:Week6; n=45, 57 | -1.7 (9.33) | 0.9 (9.38)
  SBP: Pre-Dose:Week8; n=34, 47: number analyzed (Participants) | 34 | 47
  SBP: Pre-Dose:Week8; n=34, 47 | -1.9 (7.85) | 0.4 (7.91)
  SBP: Post-DoseWeek8; n=34, 47: number analyzed (Participants) | 34 | 47
  SBP: Post-DoseWeek8; n=34, 47 | -2.7 (9.81) | 2.3 (9.46)
  SBP: Week10; n=34, 46: number analyzed (Participants) | 34 | 46
  SBP: Week10; n=34, 46 | -2.5 (10.20) | 0.7 (11.74)
  SBP: Pre-dose: Week12; n=24, 39: number analyzed (Participants) | 24 | 39
  SBP: Pre-dose: Week12; n=24, 39 | 0.3 (8.34) | 1.5 (10.19)
  SBP: Post-dose: Week12; n=24, 39: number analyzed (Participants) | 24 | 39
  SBP: Post-dose: Week12; n=24, 39 | -0.7 (6.34) | 3.3 (11.23)
  SBP: Week14; n=24, 39: number analyzed (Participants) | 24 | 39
  SBP: Week14; n=24, 39 | -1.6 (9.17) | 2.1 (10.47)
  SBP: Week16; n=24, 39: number analyzed (Participants) | 24 | 39
  SBP: Week16; n=24, 39 | -2.8 (9.16) | 1.5 (10.37)
  SBP: Week20; n=76, 78: number analyzed (Participants) | 76 | 78
  SBP: Week20; n=76, 78 | -1.0 (10.72) | 1.7 (10.32)
  SBP: Week24; n=75, 76: number analyzed (Participants) | 75 | 76
  SBP: Week24; n=75, 76 | -2.4 (10.78) | 1.7 (10.46)
  SBP: Week28; n=74, 77: number analyzed (Participants) | 74 | 77
  SBP: Week28; n=74, 77 | -1.3 (9.95) | 1.0 (9.77)
  DBP: Post-dose: Week0; n=82,83 | -0.7 (6.58) | -0.3 (5.67)
  DBP: Week1; n=79, 75: number analyzed (Participants) | 79 | 75
  DBP: Week1; n=79, 75 | 0.3 (6.96) | 0.7 (8.29)
  DBP: Week2; n=73, 75: number analyzed (Participants) | 73 | 75
  DBP: Week2; n=73, 75 | -0.7 (8.61) | -0.8 (7.04)
  DBP: Pre-dose: Week4; n=49, 59: number analyzed (Participants) | 49 | 59
  DBP: Pre-dose: Week4; n=49, 59 | -1.1 (8.26) | 0.4 (7.72)
  DBP: Post-dose: Week4; n=48, 59: number analyzed (Participants) | 48 | 59
  DBP: Post-dose: Week4; n=48, 59 | -0.4 (7.93) | 0.3 (7.79)
  DBP:Week6; n=45, 57: number analyzed (Participants) | 45 | 57
  DBP:Week6; n=45, 57 | 0.6 (7.72) | -1.0 (7.32)
  DBP: Pre-Dose:Week8; n=34, 47: number analyzed (Participants) | 34 | 47
  DBP: Pre-Dose:Week8; n=34, 47 | -0.4 (7.66) | -2.0 (7.79)
  DBP: Post-DoseWeek8; n=34, 47: number analyzed (Participants) | 34 | 47
  DBP: Post-DoseWeek8; n=34, 47 | -0.1 (7.54) | -1.2 (7.21)
  DBP: Week10; n=34, 46: number analyzed (Participants) | 34 | 46
  DBP: Week10; n=34, 46 | -0.1 (9.36) | -0.2 (7.94)
  DBP: Pre-dose: Week12; n=24, 39: number analyzed (Participants) | 24 | 39
  DBP: Pre-dose: Week12; n=24, 39 | 0.3 (7.27) | 0.6 (6.52)
  DBP: Post-dose: Week12; n=24, 39: number analyzed (Participants) | 24 | 39
  DBP: Post-dose: Week12; n=24, 39 | 0.0 (8.08) | -0.5 (6.79)
  DBP: Week14; n=24, 39: number analyzed (Participants) | 24 | 39
  DBP: Week14; n=24, 39 | 0.0 (5.28) | 0.5 (6.84)
  DBP: Week16; n=24, 39: number analyzed (Participants) | 24 | 39
  DBP: Week16; n=24, 39 | -0.3 (8.37) | -0.5 (5.59)
  DBP: Week20; n=76, 78: number analyzed (Participants) | 76 | 78
  DBP: Week20; n=76, 78 | -0.4 (8.61) | 0.7 (6.60)
  DBP: Week24; n=75, 76: number analyzed (Participants) | 75 | 76
  DBP: Week24; n=75, 76 | 0.1 (8.15) | 0.3 (7.06)
  DBP: Week28; n=74, 77: number analyzed (Participants) | 74 | 77
  DBP: Week28; n=74, 77 | -0.3 (9.74) | -0.4 (7.62)

24. Secondary Outcome: Change From Baseline in Pulse Rate (PR)
Description: Pulse rate was measured in semi-supine position after 5 minutes rest. Baseline is defined as the most recent recorded value before dosing on Day 1. Change from Baseline was calculated by subtracting Baseline value from the specified time point value. Data for change from Baseline for post dose values have been presented.
Time Frame: as for outcome 23
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 82 | 83
Beats per minute
  Post-dose: Week0; n=82, 83 | -2.2 (7.20) | -0.1 (6.54)
  Week1; n=79, 75: number analyzed (Participants) | 79 | 75
  Week1; n=79, 75 | 0.8 (6.12) | 3.1 (7.95)
  Week2; n=73, 75: number analyzed (Participants) | 73 | 75
  Week2; n=73, 75 | 2.9 (7.31) | 1.7 (7.86)
  Pre-dose:Week4; n=49, 59: number analyzed (Participants) | 49 | 59
  Pre-dose:Week4; n=49, 59 | -0.3 (9.73) | 0.1 (9.72)
  Post-dose:Week4; n=48, 59: number analyzed (Participants) | 48 | 59
  Post-dose:Week4; n=48, 59 | -2.0 (10.00) | -1.0 (10.93)
  Week6; n=45, 57: number analyzed (Participants) | 45 | 57
  Week6; n=45, 57 | 3.3 (11.85) | 2.8 (9.26)
  Pre-dose: Week8; n=34, 47: number analyzed (Participants) | 34 | 47
  Pre-dose: Week8; n=34, 47 | -0.3 (9.11) | 1.0 (7.62)
  Post-dose: Week8; n=34, 47: number analyzed (Participants) | 34 | 47
  Post-dose: Week8; n=34, 47 | -0.9 (10.39) | -0.6 (9.71)
  Week10; n=34, 46: number analyzed (Participants) | 34 | 46
  Week10; n=34, 46 | 2.6 (8.86) | 2.4 (6.72)
  Pre-dose: Week12; n=24, 39: number analyzed (Participants) | 24 | 39
  Pre-dose: Week12; n=24, 39 | 2.8 (8.04) | 1.7 (7.53)
  Post-dose: Week12; n=24, 39: number analyzed (Participants) | 24 | 39
  Post-dose: Week12; n=24, 39 | 0.9 (8.84) | -1.2 (10.57)
  Week14; n=24, 39: number analyzed (Participants) | 24 | 39
  Week14; n=24, 39 | 3.1 (9.81) | 3.6 (6.62)
  Week16; n=24, 39: number analyzed (Participants) | 24 | 39
  Week16; n=24, 39 | 3.5 (9.14) | 2.6 (8.30)
  Week20; n=76, 78: number analyzed (Participants) | 76 | 78
  Week20; n=76, 78 | 2.1 (8.34) | 3.6 (9.48)
  Week24; n=75, 76: number analyzed (Participants) | 75 | 76
  Week24; n=75, 76 | 2.3 (8.00) | 2.5 (7.98)
  Week28; n=74, 77: number analyzed (Participants) | 74 | 77
  Week28; n=74, 77 | 2.5 (8.50) | 2.3 (7.98)

25. Secondary Outcome: Change From Baseline Between Post-dose and Pre-dose in DBP and SBP
Description: DBP and SBP was measured pre-dose and post-dose in semi-supine position after 5 minutes rest. Baseline is defined as the most recent recorded value before dosing on Day 1. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline and Weeks 0, 4, 8 and 12
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 82 | 83
mmHg
  SBP: Week0; n=82, 83 | -2.0 (8.05) | 1.3 (7.19)
  SBP: Week4; n=48, 59: number analyzed (Participants) | 48 | 59
  SBP: Week4; n=48, 59 | -0.4 (5.70) | 2.4 (9.32)
  SBP: Week8; n=34, 47: number analyzed (Participants) | 34 | 47
  SBP: Week8; n=34, 47 | -0.8 (6.03) | 1.9 (6.58)
  SBP: Week12; n=24, 39: number analyzed (Participants) | 24 | 39
  SBP: Week12; n=24, 39 | -0.9 (7.51) | 1.8 (8.72)
  DBP: Week0; n=82, 83 | -0.7 (6.58) | -0.3 (5.67)
  DBP: Week4; n=48, 59: number analyzed (Participants) | 48 | 59
  DBP: Week4; n=48, 59 | 0.4 (4.95) | -0.1 (6.76)
  DBP: Week8; n=34, 47: number analyzed (Participants) | 34 | 47
  DBP: Week8; n=34, 47 | 0.2 (4.38) | 0.8 (5.55)
  DBP: Week12; n=24, 39: number analyzed (Participants) | 24 | 39
  DBP: Week12; n=24, 39 | -0.3 (4.70) | -1.1 (6.08)

26. Secondary Outcome: Change From Baseline Between Post-dose and Pre-dose in Pulse Rate
Description: Pulse rate was measured pre-dose and post-dose in semi-supine position after 5 minutes rest. Baseline is defined as the most recent recorded value before dosing on Day 1. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline and Weeks 0, 4, 8 and 12
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 82 | 83
Beats per minute
  Week0; n=82, 83 | -2.2 (7.20) | -0.1 (6.54)
  Week4; n=48, 59: number analyzed (Participants) | 48 | 59
  Week4; n=48, 59 | -1.6 (5.75) | -1.1 (6.85)
  Week8; n=34, 47: number analyzed (Participants) | 34 | 47
  Week8; n=34, 47 | -0.5 (7.21) | -1.6 (6.02)
  Week12; n=24, 39: number analyzed (Participants) | 24 | 39
  Week12; n=24, 39 | -2.0 (5.97) | -2.9 (9.05)

27. Secondary Outcome: Change From Baseline in PR Interval, QRS Duration, Uncorrected QT Interval, QT Corrected Interval-Fredericia [QTcF] Interval and RR Interval
Description: Triplicate 12-lead ECGs were recorded pre-dose and post-dose with participant in semi-supine position after 5 minutes rest. At each time point ECG was taken using an ECG machine that automatically measures PR interval, QRS duration, uncorrected QT interval, QTcF interval and RR interval. Baseline is defined as the most recent recorded value before dosing on Day 1. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline and Week 0 (Post-dose), Week 4 (Pre and Post dose), Week 8 (Pre and Post dose), Week 12 (Pre and Post dose) and Week 16
Population: Safety Population. Only those participants with data available at indicated time points were analyzed. Participants with data available at specified time points were represented by n=x in the category titles.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 80 | 80
milliseconds
  PR: Post-dose: Week0; n=80, 80 | 1.8 (9.77) | 3.1 (9.28)
  PR: Pre-dose: Week4; n=49, 59: number analyzed (Participants) | 49 | 59
  PR: Pre-dose: Week4; n=49, 59 | -0.4 (7.91) | 1.3 (10.93)
  PR: Post-dose: Week4; n=48, 59: number analyzed (Participants) | 48 | 59
  PR: Post-dose: Week4; n=48, 59 | 1.2 (9.74) | 1.9 (11.76)
  PR: Pre-dose: Week8; n=34, 47: number analyzed (Participants) | 34 | 47
  PR: Pre-dose: Week8; n=34, 47 | 0.0 (8.69) | 1.4 (11.70)
  PR:Post-dose: Week8; n=33, 47: number analyzed (Participants) | 33 | 47
  PR:Post-dose: Week8; n=33, 47 | 0.5 (11.47) | 1.5 (11.30)
  PR: Pre-dose:Week12; n=24, 39: number analyzed (Participants) | 24 | 39
  PR: Pre-dose:Week12; n=24, 39 | -1.3 (9.51) | -0.5 (13.17)
  PR: Post-dose Week12; n=24, 39: number analyzed (Participants) | 24 | 39
  PR: Post-dose Week12; n=24, 39 | 1.3 (10.85) | 2.2 (12.59)
  PR: Week16; n=24, 39: number analyzed (Participants) | 24 | 39
  PR: Week16; n=24, 39 | -0.6 (10.22) | -0.7 (12.91)
  QRS:Post-dose Week0; n=80, 80 | 0.0 (5.75) | 0.2 (5.60)
  QRS:Pre-dose Week4; n=49, 59: number analyzed (Participants) | 49 | 59
  QRS:Pre-dose Week4; n=49, 59 | -0.5 (5.69) | 0.7 (5.72)
  QRS: Post-dose:Week4; n=48, 59: number analyzed (Participants) | 48 | 59
  QRS: Post-dose:Week4; n=48, 59 | -0.2 (6.10) | 0.1 (6.14)
  QRS:Pre-dose:Week8; n=34, 47: number analyzed (Participants) | 34 | 47
  QRS:Pre-dose:Week8; n=34, 47 | 0.2 (5.86) | -0.1 (4.90)
  QRS:Post-dose:Week8; n=33, 47: number analyzed (Participants) | 33 | 47
  QRS:Post-dose:Week8; n=33, 47 | 0.5 (7.02) | 0.1 (4.87)
  QRS:Pre-dose: Week12; n=24, 39: number analyzed (Participants) | 24 | 39
  QRS:Pre-dose: Week12; n=24, 39 | -1.3 (4.83) | -1.1 (7.13)
  QRS:Post-dose: Week12; n=24, 39: number analyzed (Participants) | 24 | 39
  QRS:Post-dose: Week12; n=24, 39 | -0.7 (6.03) | -1.8 (6.21)
  QRS:Week16; n=24, 39: number analyzed (Participants) | 24 | 39
  QRS:Week16; n=24, 39 | -1.6 (6.19) | -2.0 (6.25)
  QT:Post-dose: Week0; n=80, 80 | 7.4 (19.67) | 3.5 (16.69)
  QT:Pre-dose: Week4; n=49, 59: number analyzed (Participants) | 49 | 59
  QT:Pre-dose: Week4; n=49, 59 | -1.7 (21.48) | -1.8 (17.93)
  QT:Post-dose: Week4; n=48, 59: number analyzed (Participants) | 48 | 59
  QT:Post-dose: Week4; n=48, 59 | 8.9 (23.09) | 5.1 (18.78)
  QT:Pre-dose: Week8; n=34, 47: number analyzed (Participants) | 34 | 47
  QT:Pre-dose: Week8; n=34, 47 | 3.5 (23.67) | -4.7 (20.53)
  QT:Pre-dose: Week8; n=33, 47: number analyzed (Participants) | 33 | 47
  QT:Pre-dose: Week8; n=33, 47 | 6.7 (30.69) | 7.0 (23.49)
  QT Pre-dose:Week12; n=24, 39: number analyzed (Participants) | 24 | 39
  QT Pre-dose:Week12; n=24, 39 | 1.5 (22.31) | -3.1 (23.54)
  QT:Post-dose:Week12; n=24, 39: number analyzed (Participants) | 24 | 39
  QT:Post-dose:Week12; n=24, 39 | 3.3 (24.38) | 2.4 (23.16)
  QT:Week16; n=24,39: number analyzed (Participants) | 24 | 39
  QT:Week16; n=24,39 | -2.2 (21.15) | -7.3 (20.68)
  QTcF:Post-dose:Week0; n=80, 80 | 4.2 (12.56) | 3.8 (11.21)
  QTcF:Pre-dose:Week4; n=49, 59: number analyzed (Participants) | 49 | 59
  QTcF:Pre-dose:Week4; n=49, 59 | -1.4 (11.35) | -1.0 (12.10)
  QTcF:Post-dose:Week4; n=48, 59: number analyzed (Participants) | 48 | 59
  QTcF:Post-dose:Week4; n=48, 59 | 4.0 (13.57) | 2.0 (12.46)
  QTcF:Pre-dose:Week8; n=34, 47: number analyzed (Participants) | 34 | 47
  QTcF:Pre-dose:Week8; n=34, 47 | 6.4 (13.00) | -0.9 (14.54)
  QTcF:Post-dose:Week8; n=33, 47: number analyzed (Participants) | 33 | 47
  QTcF:Post-dose:Week8; n=33, 47 | 5.5 (12.86) | 5.8 (16.08)
  QTcF:Pre-dose:Week12; n=24, 39: number analyzed (Participants) | 24 | 39
  QTcF:Pre-dose:Week12; n=24, 39 | 3.3 (13.45) | 0.4 (17.56)
  QTcF:Post-dose: Week12; n=24, 39: number analyzed (Participants) | 24 | 39
  QTcF:Post-dose: Week12; n=24, 39 | 4.4 (13.91) | 2.9 (14.33)
  QTcF: Week16; n=24, 39: number analyzed (Participants) | 24 | 39
  QTcF: Week16; n=24, 39 | -0.5 (11.87) | -2.2 (14.83)
  RR:Post-dose: Week0; n=80, 80 | 24.0 (104.42) | -0.2 (89.38)
  RR:Pre-dose: Week4; n=49, 59: number analyzed (Participants) | 49 | 59
  RR:Pre-dose: Week4; n=49, 59 | -1.3 (114.81) | -2.0 (96.20)
  RR:Post-dose: Week4; n=48, 59: number analyzed (Participants) | 48 | 59
  RR:Post-dose: Week4; n=48, 59 | 36.2 (118.51) | 26.7 (110.84)
  RR:Pre-dose:Week8; n=34, 47: number analyzed (Participants) | 34 | 47
  RR:Pre-dose:Week8; n=34, 47 | -17.4 (135.17) | -24.2 (92.65)
  RR:Post-dose:Week8; n=33, 47: number analyzed (Participants) | 33 | 47
  RR:Post-dose:Week8; n=33, 47 | 10.8 (176.36) | 10.7 (97.02)
  RR:Pre-dose:Week12; n=24, 39: number analyzed (Participants) | 24 | 39
  RR:Pre-dose:Week12; n=24, 39 | -12.6 (107.36) | -21.6 (100.97)
  RR:Post-dose:Week12; n=24, 39: number analyzed (Participants) | 24 | 39
  RR:Post-dose:Week12; n=24, 39 | -4.8 (148.89) | 1.3 (118.83)
  RR:Week16; n=24, 39: number analyzed (Participants) | 24 | 39
  RR:Week16; n=24, 39 | -14.4 (113.07) | -33.9 (102.02)

28. Secondary Outcome: Change From Baseline in ECG Heart Rate
Description: Triplicate 12-lead ECGs were recorded pre-dose and post-dose with participant in semi-supine position after 5 minutes rest. At each time point ECG was taken using an ECG machine that automatically measures heart rate. Baseline is defined as the most recent recorded value before dosing on Day 1. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: as for outcome 27
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 82 | 83
Beats per minute
  Post-dose: Week0; n=82, 83 | -1.6 (7.57) | 0.2 (6.93)
  Pre-dose: Week4; n=49, 59: number analyzed (Participants) | 49 | 59
  Pre-dose: Week4; n=49, 59 | 0.4 (9.06) | 0.7 (7.94)
  Post-dose: Week4; n=48, 59: number analyzed (Participants) | 48 | 59
  Post-dose: Week4; n=48, 59 | -2.4 (9.09) | -1.0 (8.48)
  Pre-dose: Week8; n=34, 47: number analyzed (Participants) | 34 | 47
  Pre-dose: Week8; n=34, 47 | 1.5 (11.81) | 1.9 (6.98)
  Post-dose: Week8; n=33, 47: number analyzed (Participants) | 33 | 47
  Post-dose: Week8; n=33, 47 | -0.3 (15.59) | -0.4 (7.57)
  Pre-dose:Week12; n=24, 39: number analyzed (Participants) | 24 | 39
  Pre-dose:Week12; n=24, 39 | 0.6 (8.98) | 1.6 (7.56)
  Post-dose Week12; n=24, 39: number analyzed (Participants) | 24 | 39
  Post-dose Week12; n=24, 39 | 0.4 (12.44) | 0.5 (9.28)
  Week16; n=24, 39: number analyzed (Participants) | 24 | 39
  Week16; n=24, 39 | 0.5 (10.04) | 3.1 (8.12)

29. Secondary Outcome: Change From Baseline in QRS Axis
Description: Triplicate 12-lead ECGs were recorded with participant in semi-supine position after 5 minutes rest. At each time point ECG was taken using an ECG machine that automatically measures QRS axis. Baseline is defined as the most recent recorded value before dosing on Day 1. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline and Week 4 (Pre and Post dose), Week 8 (Pre and Post dose), Week 12 (Pre and Post dose) and Week 16
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 80 | 80
Degrees
  Post-dose: Week0; n=80, 80 | -0.8 (10.76) | 1.9 (6.75)
  Pre-dose: Week4; n=49, 59: number analyzed (Participants) | 49 | 59
  Pre-dose: Week4; n=49, 59 | 0.7 (14.30) | 2.3 (13.77)
  Post-dose: Week4; n=48, 59: number analyzed (Participants) | 48 | 59
  Post-dose: Week4; n=48, 59 | -0.1 (16.72) | 1.4 (11.95)
  Pre-dose: Week8; n=34, 47: number analyzed (Participants) | 34 | 47
  Pre-dose: Week8; n=34, 47 | -0.2 (10.56) | -1.0 (9.34)
  Post-dose: Week8; n=33, 47: number analyzed (Participants) | 33 | 47
  Post-dose: Week8; n=33, 47 | 1.0 (9.88) | -1.2 (8.37)
  Pre-dose:Week12; n=24, 39: number analyzed (Participants) | 24 | 39
  Pre-dose:Week12; n=24, 39 | 0.2 (8.59) | 2.0 (31.39)
  Post-dose Week12; n=24, 39: number analyzed (Participants) | 24 | 39
  Post-dose Week12; n=24, 39 | -1.3 (9.49) | -1.2 (15.73)
  Week16; n=24, 39: number analyzed (Participants) | 24 | 39
  Week16; n=24, 39 | 2.3 (11.35) | -1.4 (10.88)

30. Secondary Outcome: Change Between Pre-dose and Post-dose of PR Interval, QRS Duration, Uncorrected QT Interval, QTcF Interval and RR Interval
Description: as for outcome 27
Time Frame: Baseline and Weeks 0, 4, 8 and 12
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 80 | 80
milliseconds
  PR:Week0; n=80, 80 | 1.8 (9.77) | 3.1 (9.28)
  PR: Week4; n=48, 59: number analyzed (Participants) | 48 | 59
  PR: Week4; n=48, 59 | 1.7 (8.04) | 0.5 (9.77)
  PR: Week8; n=33, 47: number analyzed (Participants) | 33 | 47
  PR: Week8; n=33, 47 | 0.3 (8.70) | -0.1 (9.96)
  PR: Week12; n=24, 39: number analyzed (Participants) | 24 | 39
  PR: Week12; n=24, 39 | 2.2 (10.00) | 3.0 (9.86)
  QRS:Week0; n=80, 80 | 0.0 (5.75) | 0.2 (5.60)
  QRS: Week4; n=48, 59: number analyzed (Participants) | 48 | 59
  QRS: Week4; n=48, 59 | 0.1 (4.35) | -0.8 (5.58)
  QRS:Week8; n=33, 47: number analyzed (Participants) | 33 | 47
  QRS:Week8; n=33, 47 | 0.3 (7.03) | 0.4 (4.86)
  QRS:Week12; n=24, 39: number analyzed (Participants) | 24 | 39
  QRS:Week12; n=24, 39 | 0.7 (5.36) | -0.9 (4.60)
  QT:Week0; n=80, 80 | 7.4 (19.67) | 3.5 (16.69)
  QT:Week4; n=48, 59: number analyzed (Participants) | 48 | 59
  QT:Week4; n=48, 59 | 10.8 (13.32) | 6.9 (15.63)
  QT:Week8; n=33, 47: number analyzed (Participants) | 33 | 47
  QT:Week8; n=33, 47 | 3.4 (19.22) | 11.5 (17.57)
  QT:Week12; n=24, 39: number analyzed (Participants) | 24 | 39
  QT:Week12; n=24, 39 | 1.9 (17.17) | 4.6 (18.77)
  QTcFWeek0; n=80, 80 | 4.2 (12.56) | 3.8 (11.21)
  QTcF:Week4; n=48, 59: number analyzed (Participants) | 48 | 59
  QTcF:Week4; n=48, 59 | 5.4 (9.51) | 2.9 (10.88)
  QTcF:Week8; n=33, 47: number analyzed (Participants) | 33 | 47
  QTcF:Week8; n=33, 47 | -0.7 (10.17) | 6.6 (10.65)
  QTcF:Week12; n=24, 39: number analyzed (Participants) | 24 | 39
  QTcF:Week12; n=24, 39 | 1.1 (13.28) | 2.0 (13.48)
  RR:Week0; n=80, 80 | 24.0 (104.42) | -0.2 (89.38)
  RR:Week4; n=48, 59: number analyzed (Participants) | 48 | 59
  RR:Week4; n=48, 59 | 37.6 (83.83) | 29.5 (88.38)
  RR:Week8; n=33, 47: number analyzed (Participants) | 33 | 47
  RR:Week8; n=33, 47 | 29.3 (97.67) | 34.4 (95.05)
  RR:Week12; n=24, 39: number analyzed (Participants) | 24 | 39
  RR:Week12; n=24, 39 | 8.8 (83.16) | 20.7 (104.02)

31. Secondary Outcome: Change Between Pre-dose and Post-dose of Heart Rate
Description: as for outcome 28
Time Frame: Baseline and Weeks 0, 4, 8 and 12
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 80 | 80
Beats per minute
  Week0; n=80, 80 | -1.6 (7.57) | 0.2 (6.93)
  Week4; n=48, 59: number analyzed (Participants) | 48 | 59
  Week4; n=48, 59 | -2.9 (5.79) | -1.7 (6.15)
  Week8; n=33, 47: number analyzed (Participants) | 33 | 47
  Week8; n=33, 47 | -1.8 (8.74) | -2.3 (6.83)
  Week12; n=24, 39: number analyzed (Participants) | 24 | 39
  Week12; n=24, 39 | -0.2 (6.69) | -0.9 (7.75)

32. Secondary Outcome: Change Between Pre-dose and Post-dose of QRS Axis
Description: Triplicate 12-lead ECGs were recorded pre-dose and post-dose with participant in semi-supine position after 5 minutes rest. At each time point ECG was taken using an ECG machine that automatically measures QRS axis. Baseline is defined as the most recent recorded value before dosing on Day 1. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline and Weeks 0, 4, 8 and 12
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 80 | 80
Degrees
  Week0; n=80, 80 | -0.8 (10.76) | 1.9 (6.75)
  Week4; n=48, 59: number analyzed (Participants) | 48 | 59
  Week4; n=48, 59 | -0.3 (9.20) | -0.9 (16.22)
  Week8; n=33, 47: number analyzed (Participants) | 33 | 47
  Week8; n=33, 47 | 1.2 (10.01) | -0.2 (9.30)
  Week12; n=24, 39: number analyzed (Participants) | 24 | 39
  Week12; n=24, 39 | -1.6 (6.44) | 2.8 (14.25)

33. Secondary Outcome: Change From Baseline in Maximum, Minimum and Average Changes in Heart Rate
Description: Using a Holter monitor, maximum, minimum and average changes in heart rate was recorded at Baseline, Weeks 0, 4 and 12 through 24 hours. Participants with analyzable time of at least 16 hours were evaluated. Baseline is the value from the screening visit assessment. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline and Weeks 0, 4 and 12
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 81 | 80
Beats per minute
  Mean Heart Rate: Week0; n=81, 80 | -1.1 (6.56) | -2.0 (6.00)
  Mean Heart Rate: Week4; n=49, 58: number analyzed (Participants) | 49 | 58
  Mean Heart Rate: Week4; n=49, 58 | 76.8 (10.60) | 80.0 (10.80)
  Mean Heart Rate: Week12; n=24, 37: number analyzed (Participants) | 24 | 37
  Mean Heart Rate: Week12; n=24, 37 | 78.8 (11.12) | 79.9 (10.08)
  Maximum Heart Rate: Week0; n=81, 80 | -0.3 (13.13) | -5.0 (14.55)
  Maximum Heart Rate: Week4; n=49, 58: number analyzed (Participants) | 49 | 58
  Maximum Heart Rate: Week4; n=49, 58 | 128.3 (13.03) | 130.3 (16.41)
  Maximum Heart Rate: Week12; n=24, 37: number analyzed (Participants) | 24 | 37
  Maximum Heart Rate: Week12; n=24, 37 | 128.5 (15.21) | 132.1 (15.80)
  Minimum Heart Rate: Week0; n=81, 80 | -0.8 (5.08) | -0.8 (4.55)
  Minimum Heart Rate: Week4; n=49, 58: number analyzed (Participants) | 49 | 58
  Minimum Heart Rate: Week4; n=49, 58 | 50.6 (7.49) | 53.8 (8.15)
  Minimum Heart Rate: Week12; n=24, 37: number analyzed (Participants) | 24 | 37
  Minimum Heart Rate: Week12; n=24, 37 | 53.6 (7.49) | 53.4 (9.09)

34. Secondary Outcome: Change From Baseline in Supraventricular Couplets, Supraventricular Ectopics, Supraventricular Runs, Supraventricular Singles, Ventricular Couplets, Ventricular Ectopics, Ventricular Runs, Ventricular Singles
Description: Using a Holter monitor, supraventricular couplets, supraventricular ectopics, supraventricular runs, supraventricular singles, ventricular couplets, ventricular ectopics, ventricular runs, ventricular singles were recorded at Baseline, Weeks 0, 4 and 12 through 24 hours. Participants with analyzable time of at least 16 hours were evaluated. Baseline is the value from the screening visit assessment. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline and Weeks 0, 4 and 12
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Events per hour
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 81 | 80
Events per hour
  supraventricular couplets: Week0; n=81, 80 | -2.0 (21.68) | 16.5 (144.04)
  supraventricular couplets: Week4; n=49, 58: number analyzed (Participants) | 49 | 58
  supraventricular couplets: Week4; n=49, 58 | -1.9 (14.11) | -2.2 (9.86)
  supraventricular couplets: Week12; n=24, 37: number analyzed (Participants) | 24 | 37
  supraventricular couplets: Week12; n=24, 37 | -3.9 (35.82) | -0.5 (3.48)
  supraventricular ectopics: Week0; n=81, 80 | 2.6 (369.71) | 6.8 (188.46)
  supraventricular ectopics: Week4; n=49, 58: number analyzed (Participants) | 49 | 58
  supraventricular ectopics: Week4; n=49, 58 | -30.9 (445.93) | -7.3 (148.20)
  supraventricular ectopics: Week12; n=24, 37: number analyzed (Participants) | 24 | 37
  supraventricular ectopics: Week12; n=24, 37 | 34.9 (300.07) | 9.4 (94.82)
  supraventricular runs: Week0; n=81, 80 | -0.5 (3.62) | 0.2 (2.09)
  supraventricular runs: Week4; n=49, 58: number analyzed (Participants) | 49 | 58
  supraventricular runs: Week4; n=49, 58 | -0.1 (2.37) | -0.6 (3.01)
  supraventricular runs: Week12; n=24, 37: number analyzed (Participants) | 24 | 37
  supraventricular runs: Week12; n=24, 37 | -1.1 (6.30) | -0.4 (1.83)
  supraventricular singles: Week0; n=81, 80 | 9.0 (349.81) | -13.1 (120.73)
  supraventricular singles: Week4; n=49, 58: number analyzed (Participants) | 49 | 58
  supraventricular singles: Week4; n=49, 58 | -25.3 (425.20) | -3.1 (138.30)
  supraventricular singles: Week12; n=24, 37: number analyzed (Participants) | 24 | 37
  supraventricular singles: Week12; n=24, 37 | 45.5 (263.03) | 8.4 (89.64)
  ventricular couplets: Week0; n=81, 80 | 0.7 (3.80) | -0.1 (1.59)
  ventricular couplets: Week4; n=49, 58: number analyzed (Participants) | 49 | 58
  ventricular couplets: Week4; n=49, 58 | 0.2 (0.80) | 0.1 (0.65)
  ventricular couplets: Week12; n=24, 37: number analyzed (Participants) | 24 | 37
  ventricular couplets: Week12; n=24, 37 | 0.0 (0.00) | 0.3 (1.43)
  ventricular ectopics: Week0; n=81, 80 | 44.6 (265.28) | -12.2 (141.39)
  ventricular ectopics: Week4; n=49, 58: number analyzed (Participants) | 49 | 58
  ventricular ectopics: Week4; n=49, 58 | -10.7 (105.24) | 6.4 (54.80)
  ventricular ectopics: Week12; n=24, 37: number analyzed (Participants) | 24 | 37
  ventricular ectopics: Week12; n=24, 37 | -5.3 (52.78) | 176.0 (926.75)
  ventricular runs: Week0; n=81, 80 | 0.0 (0.25) | 0.0 (0.19)
  ventricular runs: Week4; n=49, 58: number analyzed (Participants) | 49 | 58
  ventricular runs: Week4; n=49, 58 | 0.0 (0.29) | 0.0 (0.00)
  ventricular runs: Week12; n=24, 37: number analyzed (Participants) | 24 | 37
  ventricular runs: Week12; n=24, 37 | 0.0 (0.29) | 0.0 (0.00)
  ventricular singles: Week0; n=81, 80 | 44.0 (228.09) | -12.2 (139.28)
  ventricular singles: Week4; n=49, 58: number analyzed (Participants) | 49 | 58
  ventricular singles: Week4; n=49, 58 | -10.4 (104.12) | 6.3 (53.79)
  ventricular singles: Week12; n=24, 37: number analyzed (Participants) | 24 | 37
  ventricular singles: Week12; n=24, 37 | -5.4 (53.23) | 174.5 (921.42)

35. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter: Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP), Gamma- Glutamyl Transferase (GGT) and Creatine Kinase (CK)
Description: Blood samples were collected for the analysis of clinical chemistry parameters including AST, ALT, ALP, GGT and CK at indicated time points. Baseline is defined as the most recent recorded value before dosing on Day 1. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16 and 28
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 74 | 74
International units per liter
  ALT: Week 2; n=72, 74: number analyzed (Participants) | 72 | 74
  ALT: Week 2; n=72, 74 | -0.9 (8.88) | -0.2 (7.07)
  ALT:Week 4; n=47,59: number analyzed (Participants) | 47 | 59
  ALT:Week 4; n=47,59 | -0.5 (9.50) | -2.6 (7.24)
  ALT: Week 8; n=34,47: number analyzed (Participants) | 34 | 47
  ALT: Week 8; n=34,47 | -0.1 (6.93) | -2.4 (7.30)
  ALT: Week 12; n=24, 36: number analyzed (Participants) | 24 | 36
  ALT: Week 12; n=24, 36 | -1.6 (6.86) | -2.4 (7.77)
  ALT: Week 16; n=24, 39: number analyzed (Participants) | 24 | 39
  ALT: Week 16; n=24, 39 | -1.2 (7.97) | -2.6 (6.54)
  ALT: Week 28; n=74, 74 | -1.1 (9.57) | -0.9 (10.51)
  ALP: Week 2; n=72, 74: number analyzed (Participants) | 72 | 74
  ALP: Week 2; n=72, 74 | -1.9 (8.32) | -0.8 (8.96)
  ALP:Week 4; n=47, 59: number analyzed (Participants) | 47 | 59
  ALP:Week 4; n=47, 59 | -0.8 (13.18) | -1.0 (8.17)
  ALP:Week 8; n=34, 47: number analyzed (Participants) | 34 | 47
  ALP:Week 8; n=34, 47 | 0.9 (7.37) | -2.3 (8.64)
  ALP:Week 12; n =24, 36: number analyzed (Participants) | 24 | 36
  ALP:Week 12; n =24, 36 | 2.4 (8.79) | -3.0 (14.01)
  ALP:Week 16; n=24, 39: number analyzed (Participants) | 24 | 39
  ALP:Week 16; n=24, 39 | 1.0 (9.33) | -2.3 (9.75)
  ALP:Week 28; n=74, 74 | -0.4 (12.33) | -1.2 (13.25)
  AST: Week 2; n=72, 74: number analyzed (Participants) | 72 | 74
  AST: Week 2; n=72, 74 | -0.8 (9.30) | -1.5 (6.59)
  AST:Week 4; n=47,59: number analyzed (Participants) | 47 | 59
  AST:Week 4; n=47,59 | -1.0 (6.02) | -2.5 (6.75)
  AST:Week 8, n=34,47: number analyzed (Participants) | 34 | 47
  AST:Week 8, n=34,47 | -1.6 (6.58) | -2.7 (6.36)
  AST:Week 12, n=24, 36: number analyzed (Participants) | 24 | 36
  AST:Week 12, n=24, 36 | -1.8 (4.91) | -4.1 (6.59)
  AST:Week 16, n=24, 39: number analyzed (Participants) | 24 | 39
  AST:Week 16, n=24, 39 | -1.4 (6.01) | -3.3 (6.70)
  AST:Week 28, n=74, 74 | -2.3 (6.96) | -1.7 (8.64)
  CK: Week 2, n=72, 74: number analyzed (Participants) | 72 | 74
  CK: Week 2, n=72, 74 | -12.5 (92.00) | -18.8 (207.72)
  CK:Week 4, n=47,59: number analyzed (Participants) | 47 | 59
  CK:Week 4, n=47,59 | -30.3 (68.86) | -45.1 (231.07)
  CK:Week 8, n=34,47: number analyzed (Participants) | 34 | 47
  CK:Week 8, n=34,47 | -26.6 (57.01) | -32.9 (242.98)
  CK:Week 12, n=24, 36: number analyzed (Participants) | 24 | 36
  CK:Week 12, n=24, 36 | -5.0 (73.56) | -54.5 (282.17)
  CK:Week 16, n=24, 39: number analyzed (Participants) | 24 | 39
  CK:Week 16, n=24, 39 | -20.8 (81.02) | -46.8 (272.08)
  CK:Week 28, n=74, 74 | -8.5 (131.56) | -30.7 (199.41)
  GGT: Week 2, n=72, 74: number analyzed (Participants) | 72 | 74
  GGT: Week 2, n=72, 74 | -3.2 (9.61) | -1.2 (12.16)
  GGT:Week 4, n=47,59: number analyzed (Participants) | 47 | 59
  GGT:Week 4, n=47,59 | -3.9 (14.00) | -2.5 (21.35)
  GGT:Week 8, n=34,47: number analyzed (Participants) | 34 | 47
  GGT:Week 8, n=34,47 | -3.5 (13.50) | -2.8 (15.61)
  GGT:Week 12, 24, 36: number analyzed (Participants) | 24 | 36
  GGT:Week 12, 24, 36 | -0.3 (5.87) | -5.4 (19.48)
  GGT:Week 16, n=24, 39: number analyzed (Participants) | 24 | 39
  GGT:Week 16, n=24, 39 | -1.1 (4.41) | -3.9 (14.64)
  GGT:Week 28, n=74, 73: number analyzed (Participants) | 74 | 73
  GGT:Week 28, n=74, 73 | -3.2 (13.80) | -0.7 (16.06)

36. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Glucose, Potassium, Sodium, Calcium, Phosphate, Chloride, Urea and Carbon Dioxide (CO2)
Description: Blood samples were collected at given time points to assess clinical chemistry parameters including glucose, potassium, sodium, calcium, Phosphate, chloride, urea and CO2 levels. Baseline is defined as the most recent recorded value before dosing on Day 1. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16 and 28
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 74 | 74
Millimoles per liter
  Glucose: Week 2; n=72, 74: number analyzed (Participants) | 72 | 74
  Glucose: Week 2; n=72, 74 | 0.13 (0.996) | 0.05 (1.273)
  Glucose:Week 4; n=47,59: number analyzed (Participants) | 47 | 59
  Glucose:Week 4; n=47,59 | 0.18 (0.784) | 0.19 (1.156)
  Glucose:Week 8; n=34,47: number analyzed (Participants) | 34 | 47
  Glucose:Week 8; n=34,47 | 0.26 (1.008) | 0.00 (1.400)
  Glucose:Week 12; n=24, 36: number analyzed (Participants) | 24 | 36
  Glucose:Week 12; n=24, 36 | -0.04 (0.796) | 0.20 (1.516)
  Glucose:Week 16; n=24, 39: number analyzed (Participants) | 24 | 39
  Glucose:Week 16; n=24, 39 | -0.10 (1.057) | 0.12 (0.984)
  Glucose:Week 28; n=74, 73: number analyzed (Participants) | 74 | 73
  Glucose:Week 28; n=74, 73 | 0.30 (1.245) | 0.04 (1.780)
  Potassium: Week 2; n=72, 74: number analyzed (Participants) | 72 | 74
  Potassium: Week 2; n=72, 74 | 0.14 (0.366) | 0.13 (0.596)
  Potassium:Week 4; n=47,59: number analyzed (Participants) | 47 | 59
  Potassium:Week 4; n=47,59 | 0.04 (0.361) | 0.05 (0.402)
  Potassium:Week 8; n=34,47: number analyzed (Participants) | 34 | 47
  Potassium:Week 8; n=34,47 | -0.01 (0.352) | -0.04 (0.397)
  Potassium:Week 12; n=24, 36: number analyzed (Participants) | 24 | 36
  Potassium:Week 12; n=24, 36 | 0.02 (0.363) | 0.00 (0.439)
  Potassium:Week 16; n=24, 39: number analyzed (Participants) | 24 | 39
  Potassium:Week 16; n=24, 39 | -0.09 (0.403) | 0.00 (0.439)
  Potassium:Week 28; n=74, 73: number analyzed (Participants) | 74 | 73
  Potassium:Week 28; n=74, 73 | 0.01 (0.407) | 0.01 (0.416)
  Sodium: Week 2; n=72, 74: number analyzed (Participants) | 72 | 74
  Sodium: Week 2; n=72, 74 | 0.3 (2.19) | -0.1 (2.31)
  Sodium:Week 4; n=47,59: number analyzed (Participants) | 47 | 59
  Sodium:Week 4; n=47,59 | 0.0 (1.65) | -0.9 (2.34)
  Sodium:Week 8; n=34,47: number analyzed (Participants) | 34 | 47
  Sodium:Week 8; n=34,47 | -0.1 (1.41) | -0.6 (1.51)
  Sodium:Week 12; n=24, 36: number analyzed (Participants) | 24 | 36
  Sodium:Week 12; n=24, 36 | -0.3 (2.17) | -1.1 (1.71)
  Sodium:Week 16; n=24, 39: number analyzed (Participants) | 24 | 39
  Sodium:Week 16; n=24, 39 | -0.2 (2.14) | -0.3 (2.01)
  Sodium:Week 28; n=74, 73: number analyzed (Participants) | 74 | 73
  Sodium:Week 28; n=74, 73 | 0.5 (2.55) | -0.2 (2.11)
  Calcium: Week 2; n=72, 74: number analyzed (Participants) | 72 | 74
  Calcium: Week 2; n=72, 74 | -0.006 (0.0691) | 0.001 (0.0925)
  Calcium:Week 4; n=47,59: number analyzed (Participants) | 47 | 59
  Calcium:Week 4; n=47,59 | -0.013 (0.0873) | -0.005 (0.0743)
  Calcium:Week 8; n=34,47: number analyzed (Participants) | 34 | 47
  Calcium:Week 8; n=34,47 | -0.005 (0.0648) | -0.003 (0.0997)
  Calcium:Week 12; n=24, 36: number analyzed (Participants) | 24 | 36
  Calcium:Week 12; n=24, 36 | 0.018 (0.0962) | -0.004 (0.0949)
  Calcium:Week 16; n=24, 39: number analyzed (Participants) | 24 | 39
  Calcium:Week 16; n=24, 39 | 0.014 (0.0950) | 0.017 (0.0963)
  Calcium:Week 28; n=74, 73: number analyzed (Participants) | 74 | 73
  Calcium:Week 28; n=74, 73 | 0.001 (0.0776) | 0.001 (0.0994)
  Phosphate: Week 2; n=72, 74: number analyzed (Participants) | 72 | 74
  Phosphate: Week 2; n=72, 74 | 0.031 (0.1467) | -0.023 (0.1502)
  Phosphate:Week 4; n=47,59: number analyzed (Participants) | 47 | 59
  Phosphate:Week 4; n=47,59 | 0.003 (0.1312) | -0.011 (0.1362)
  Phosphate:Week 8; n=34,47: number analyzed (Participants) | 34 | 47
  Phosphate:Week 8; n=34,47 | 0.006 (0.1678) | -0.049 (0.1420)
  Phosphate:Week 12; n=24, 36: number analyzed (Participants) | 24 | 36
  Phosphate:Week 12; n=24, 36 | 0.025 (0.1133) | -0.013 (0.1495)
  Phosphate:Week 16; n=24, 39: number analyzed (Participants) | 24 | 39
  Phosphate:Week 16; n=24, 39 | -0.006 (0.1370) | -0.019 (0.1503)
  Phosphate:Week 28; n=74, 73: number analyzed (Participants) | 74 | 73
  Phosphate:Week 28; n=74, 73 | -0.013 (0.1854) | -0.018 (0.1743)
  Chloride: Week 2; n=72, 74: number analyzed (Participants) | 72 | 74
  Chloride: Week 2; n=72, 74 | 0.3 (2.47) | 0.1 (2.22)
  Chloride:Week 4; n=47,59: number analyzed (Participants) | 47 | 59
  Chloride:Week 4; n=47,59 | 0.0 (2.04) | -0.3 (2.18)
  Chloride:Week 8; n=34,47: number analyzed (Participants) | 34 | 47
  Chloride:Week 8; n=34,47 | -0.2 (1.97) | 0.0 (2.03)
  Chloride:Week 12; n=24, 36: number analyzed (Participants) | 24 | 36
  Chloride:Week 12; n=24, 36 | -0.1 (2.61) | -0.3 (2.13)
  Chloride:Week 16; n=24, 39: number analyzed (Participants) | 24 | 39
  Chloride:Week 16; n=24, 39 | -0.4 (2.95) | -0.2 (2.61)
  Chloride:Week 28; n=74, 73: number analyzed (Participants) | 74 | 73
  Chloride:Week 28; n=74, 73 | 0.6 (2.65) | 0.7 (2.24)
  CO2: Week 2; n=72, 74: number analyzed (Participants) | 72 | 74
  CO2: Week 2; n=72, 74 | -0.4 (2.71) | 0.4 (2.10)
  CO2:Week 4; n=47,59: number analyzed (Participants) | 47 | 59
  CO2:Week 4; n=47,59 | -0.4 (2.26) | 0.3 (2.82)
  CO2:Week 8; n=34,46: number analyzed (Participants) | 34 | 46
  CO2:Week 8; n=34,46 | -0.3 (1.95) | -0.3 (1.84)
  CO2:Week 12; n=24, 36: number analyzed (Participants) | 24 | 36
  CO2:Week 12; n=24, 36 | -0.5 (2.60) | -0.1 (2.10)
  CO2:Week 16; n=24, 39: number analyzed (Participants) | 24 | 39
  CO2:Week 16; n=24, 39 | -0.5 (2.34) | 0.1 (2.28)
  CO2:Week 28; n=74, 73: number analyzed (Participants) | 74 | 73
  CO2:Week 28; n=74, 73 | -0.1 (2.28) | 0.3 (2.15)
  Urea: Week 2; n=72, 74: number analyzed (Participants) | 72 | 74
  Urea: Week 2; n=72, 74 | 0.08 (1.311) | -0.14 (1.108)
  Urea:Week 4; n=47,59: number analyzed (Participants) | 47 | 59
  Urea:Week 4; n=47,59 | 0.16 (1.344) | -0.14 (1.102)
  Urea:Week 8; n=34,47: number analyzed (Participants) | 34 | 47
  Urea:Week 8; n=34,47 | -0.04 (1.264) | 0.27 (1.151)
  Urea:Week 12; n=24, 36: number analyzed (Participants) | 24 | 36
  Urea:Week 12; n=24, 36 | 0.58 (1.537) | -0.06 (1.346)
  Urea:Week 16; n=24, 39: number analyzed (Participants) | 24 | 39
  Urea:Week 16; n=24, 39 | 0.48 (1.379) | 0.03 (1.287)
  Urea:Week 28; n=74, 73: number analyzed (Participants) | 74 | 73
  Urea:Week 28; n=74, 73 | 0.08 (1.089) | 0.16 (1.121)

37. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Creatinine, Total Bilirubin and Direct Bilirubin
Description: Blood samples were collected for the analysis of clinical chemistry parameters including total bilirubin, creatinine and direct bilirubin at indicated time points. Baseline is defined as the most recent recorded value before dosing on Day 1. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16 and 28
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 74 | 74
Micromoles per liter
  Creatinine: Week 2; n=72, 74: number analyzed (Participants) | 72 | 74
  Creatinine: Week 2; n=72, 74 | 2.35 (6.911) | 1.71 (8.321)
  Creatinine:Week 4; n=47, 59: number analyzed (Participants) | 47 | 59
  Creatinine:Week 4; n=47, 59 | 2.35 (8.319) | 0.72 (6.610)
  Creatinine:Week 8; n=34, 47: number analyzed (Participants) | 34 | 47
  Creatinine:Week 8; n=34, 47 | 1.18 (7.677) | 1.76 (6.072)
  Creatinine:Week 12; n=24, 36: number analyzed (Participants) | 24 | 36
  Creatinine:Week 12; n=24, 36 | 2.42 (6.521) | 0.02 (5.866)
  Creatinine:Week 16; n=24, 39: number analyzed (Participants) | 24 | 39
  Creatinine:Week 16; n=24, 39 | 2.50 (8.685) | 0.91 (6.105)
  Creatinine:Week 28; n=74, 73: number analyzed (Participants) | 74 | 73
  Creatinine:Week 28; n=74, 73 | 4.32 (6.810) | 2.9 (6.356)
  Total Bilirubin : Week 2; n=72, 74: number analyzed (Participants) | 72 | 74
  Total Bilirubin : Week 2; n=72, 74 | -0.1 (3.22) | 0.1 (2.83)
  Total Bilirubin :Week 4; n=47, 59: number analyzed (Participants) | 47 | 59
  Total Bilirubin :Week 4; n=47, 59 | -0.3 (3.24) | -0.4 (2.98)
  Total Bilirubin :Week 8; n=34, 47: number analyzed (Participants) | 34 | 47
  Total Bilirubin :Week 8; n=34, 47 | -0.1 (2.46) | -0.2 (4.04)
  Total Bilirubin :Week 12; n=24, 36: number analyzed (Participants) | 24 | 36
  Total Bilirubin :Week 12; n=24, 36 | -0.6 (2.32) | 0.1 (4.56)
  Total Bilirubin :Week 16; n=24, 39: number analyzed (Participants) | 24 | 39
  Total Bilirubin :Week 16; n=24, 39 | 0.0 (2.83) | -0.3 (3.39)
  Total Bilirubin :Week 28; n=74, 74 | 0.1 (2.77) | -0.5 (3.94)
  Direct bilirubin : Week 2; n=72, 74: number analyzed (Participants) | 72 | 74
  Direct bilirubin : Week 2; n=72, 74 | -0.1 (1.18) | 0.0 (1.02)
  Direct bilirubin :Week 4; n=47,59: number analyzed (Participants) | 47 | 59
  Direct bilirubin :Week 4; n=47,59 | -0.1 (0.97) | 0.1 (1.11)
  Direct bilirubin :Week 8; n=34, 47: number analyzed (Participants) | 34 | 47
  Direct bilirubin :Week 8; n=34, 47 | -0.1 (1.04) | 0.2 (1.17)
  Direct bilirubin :Week 12; n=24, 36: number analyzed (Participants) | 24 | 36
  Direct bilirubin :Week 12; n=24, 36 | -0.4 (1.18) | 0.2 (1.11)
  Direct bilirubin :Week 16; n=24, 39: number analyzed (Participants) | 24 | 39
  Direct bilirubin :Week 16; n=24, 39 | 0.1 (1.50) | 0.1 (1.07)
  Direct bilirubin :Week 28; n=74, 74 | 0.1 (1.17) | 0.1 (1.13)

38. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Total Protein and Albumin
Description: Blood samples were collected at given time points to assess clinical chemistry parameters including total protein and albumin levels. Baseline is defined as the most recent recorded value before dosing on Day 1. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16 and 28
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 74 | 74
Grams per liter
  Total Protein: Week 2, n=72, 74: number analyzed (Participants) | 72 | 74
  Total Protein: Week 2, n=72, 74 | -0.5 (3.49) | 0.4 (3.71)
  Total Protein:Week 4, n=47,59: number analyzed (Participants) | 47 | 59
  Total Protein:Week 4, n=47,59 | -0.4 (3.44) | -0.4 (3.76)
  Total Protein:Week 8, n=34,47: number analyzed (Participants) | 34 | 47
  Total Protein:Week 8, n=34,47 | 0.1 (3.20) | 0.8 (3.83)
  Total Protein:Week 12, n=24, 36: number analyzed (Participants) | 24 | 36
  Total Protein:Week 12, n=24, 36 | 0.2 (4.05) | -0.6 (4.79)
  Total Protein:Week 16, n=24, 39: number analyzed (Participants) | 24 | 39
  Total Protein:Week 16, n=24, 39 | 0.5 (4.33) | 0.4 (3.34)
  Total Protein:Week 28, n=74, 73: number analyzed (Participants) | 74 | 73
  Total Protein:Week 28, n=74, 73 | -0.8 (4.04) | -0.2 (4.27)
  Albumin: Week 2, n=72, 74: number analyzed (Participants) | 72 | 74
  Albumin: Week 2, n=72, 74 | -0.5 (2.38) | -0.4 (2.11)
  Albumin:Week 4, n=47,59: number analyzed (Participants) | 47 | 59
  Albumin:Week 4, n=47,59 | -0.5 (2.29) | -0.8 (2.62)
  Albumin:Week 8, n=34,47: number analyzed (Participants) | 34 | 47
  Albumin:Week 8, n=34,47 | -0.4 (2.36) | 0.0 (2.38)
  Albumin:Week 12, n=24, 36: number analyzed (Participants) | 24 | 36
  Albumin:Week 12, n=24, 36 | -0.3 (2.40) | -0.9 (2.69)
  Albumin:Week 16, n=24, 39: number analyzed (Participants) | 24 | 39
  Albumin:Week 16, n=24, 39 | -0.1 (2.82) | -0.4 (2.25)
  Albumin:Week 28, n=74, 73: number analyzed (Participants) | 74 | 73
  Albumin:Week 28, n=74, 73 | -0.6 (2.70) | -0.6 (2.99)

39. Secondary Outcome: Change From Baseline in Hematology Parameters: Basophil, Eosinophils, Leukocytes, Lymphocytes, Neutrophils, Monocytes, and Platelets
Description: Blood samples were collected at given time points to assess hematology parameters including basophil, eosinophils, leukocytes, lymphocytes, leutrophils, monocytes, and platelets . Baseline is defined as the most recent recorded value before dosing on Day 1. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline and Weeks1, 2, 4, 6, 8, 10, 12, 14, 16 and 28
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 78 | 74
10^9 cells per liter
  Basophil: Week 1; n=77, 74: number analyzed (Participants) | 77 | 74
  Basophil: Week 1; n=77, 74 | 0.001 (0.0361) | -0.001 (0.0396)
  Basophil:Week 2; n= 68, 72: number analyzed (Participants) | 68 | 72
  Basophil:Week 2; n= 68, 72 | 0.003 (0.0350) | 0.005 (0.0346)
  Basophil:Week 4; n=48, 57: number analyzed (Participants) | 48 | 57
  Basophil:Week 4; n=48, 57 | 0.005 (0.0341) | 0.004 (0.0409)
  Basophil:Week 6; n=43, 54: number analyzed (Participants) | 43 | 54
  Basophil:Week 6; n=43, 54 | 0.006 (0.0420) | 0.007 (0.0363)
  Basophil:Week 8; n=33, 46: number analyzed (Participants) | 33 | 46
  Basophil:Week 8; n=33, 46 | 0.002 (0.0449) | -0.001 (0.0366)
  Basophil:Week 10; n= 32, 44: number analyzed (Participants) | 32 | 44
  Basophil:Week 10; n= 32, 44 | 0.004 (0.0345) | 0.010 (0.0367)
  Basophil:Week 12; n=24, 39: number analyzed (Participants) | 24 | 39
  Basophil:Week 12; n=24, 39 | 0.010 (0.0262) | 0.010 (0.0312)
  Basophil:Week 14; n=23, 39: number analyzed (Participants) | 23 | 39
  Basophil:Week 14; n=23, 39 | -0.003 (0.0255) | 0.012 (0.0338)
  Basophil:Week 16; n=23, 39: number analyzed (Participants) | 23 | 39
  Basophil:Week 16; n=23, 39 | -0.005 (0.0316) | 0.006 (0.0409)
  Basophil:Week 28; n= 65, 60: number analyzed (Participants) | 65 | 60
  Basophil:Week 28; n= 65, 60 | 0.006 (0.0364) | 0.007 (0.0353)
  Eosinophil: Week 1; n=77, 74: number analyzed (Participants) | 77 | 74
  Eosinophil: Week 1; n=77, 74 | -0.031 (0.2868) | -0.038 (0.1424)
  Eosinophil:Week 2; n=68, 72: number analyzed (Participants) | 68 | 72
  Eosinophil:Week 2; n=68, 72 | -0.050 (0.2105) | -0.051 (0.1892)
  Eosinophil:Week 4; n=48, 57: number analyzed (Participants) | 48 | 57
  Eosinophil:Week 4; n=48, 57 | -0.048 (0.2585) | -0.119 (0.1522)
  Eosinophil:Week 6; n =43, 54: number analyzed (Participants) | 43 | 54
  Eosinophil:Week 6; n =43, 54 | -0.023 (0.2714) | -0.119 (0.1950)
  Eosinophil:Week 8; n= 33, 46: number analyzed (Participants) | 33 | 46
  Eosinophil:Week 8; n= 33, 46 | -0.014 (0.2069) | -0.096 (0.2134)
  Eosinophil:Week 10 n=32, 44: number analyzed (Participants) | 32 | 44
  Eosinophil:Week 10 n=32, 44 | 0.000 (0.2387) | -0.041 (0.2371)
  Eosinophil:Week 12; n=24, 39: number analyzed (Participants) | 24 | 39
  Eosinophil:Week 12; n=24, 39 | -0.039 (0.2621) | -0.066 (0.1939)
  Eosinophil:Week 14; n=23, 39: number analyzed (Participants) | 23 | 39
  Eosinophil:Week 14; n=23, 39 | 0.018 (0.1888) | -0.034 (0.2481)
  Eosinophil:Week 16; n=23, 39: number analyzed (Participants) | 23 | 39
  Eosinophil:Week 16; n=23, 39 | -0.018 (0.2456) | -0.093 (0.2350)
  Eosinophil:Week 28; n= 65, 60: number analyzed (Participants) | 65 | 60
  Eosinophil:Week 28; n= 65, 60 | 0.010 (0.2077) | -0.087 (0.1865)
  Leukocytes: Week 1; n=78, 74 | 0.14 (1.614) | 0.07 (1.314)
  Leukocytes:Week 2; n= 68, 73: number analyzed (Participants) | 68 | 73
  Leukocytes:Week 2; n= 68, 73 | 0.01 (1.202) | 0.09 (1.117)
  Leukocytes:Week 4; n =48, 57: number analyzed (Participants) | 48 | 57
  Leukocytes:Week 4; n =48, 57 | 0.24 (1.406) | 0.19 (1.401)
  Leukocytes:Week 6; n=43, 54: number analyzed (Participants) | 43 | 54
  Leukocytes:Week 6; n=43, 54 | 0.37 (1.346) | -0.12 (1.040)
  Leukocytes:Week 8; n=33, 47: number analyzed (Participants) | 33 | 47
  Leukocytes:Week 8; n=33, 47 | 0.08 (1.045) | 0.14 (2.248)
  Leukocytes:Week 10; n=33, 45: number analyzed (Participants) | 33 | 45
  Leukocytes:Week 10; n=33, 45 | 0.01 (1.102) | 0.03 (1.259)
  Leukocytes:Week 12; n=24, 39: number analyzed (Participants) | 24 | 39
  Leukocytes:Week 12; n=24, 39 | 0.13 (1.257) | 0.18 (1.038)
  Leukocytes:Week 14; n= 23, 39: number analyzed (Participants) | 23 | 39
  Leukocytes:Week 14; n= 23, 39 | -0.17 (1.324) | 0.26 (1.220)
  Leukocytes:Week 16; n=23, 39: number analyzed (Participants) | 23 | 39
  Leukocytes:Week 16; n=23, 39 | -0.41 (1.296) | 0.18 (1.511)
  Leukocytes:Week 28; n=65, 63: number analyzed (Participants) | 65 | 63
  Leukocytes:Week 28; n=65, 63 | -0.08 (1.545) | 0.09 (1.392)
  Lymphocytes: Week 1; n=77, 74: number analyzed (Participants) | 77 | 74
  Lymphocytes: Week 1; n=77, 74 | 0.036 (0.4248) | -0.008 (0.3292)
  Lymphocytes:Week 2; n=68, 72: number analyzed (Participants) | 68 | 72
  Lymphocytes:Week 2; n=68, 72 | 0.006 (0.3437) | 0.039 (0.4112)
  Lymphocytes:Week 4; n=48, 57: number analyzed (Participants) | 48 | 57
  Lymphocytes:Week 4; n=48, 57 | 0.043 (0.4048) | 0.061 (0.2995)
  Lymphocytes:Week 6; n=43, 54: number analyzed (Participants) | 43 | 54
  Lymphocytes:Week 6; n=43, 54 | 0.140 (0.4994) | 0.086 (0.3986)
  Lymphocytes:Week 8; n=33, 46: number analyzed (Participants) | 33 | 46
  Lymphocytes:Week 8; n=33, 46 | 0.132 (0.3257) | 0.033 (0.3477)
  Lymphocytes:Week 10; n=32, 44: number analyzed (Participants) | 32 | 44
  Lymphocytes:Week 10; n=32, 44 | 0.103 (0.4275) | 0.105 (0.4105)
  Lymphocytes:Week 12; n=24, 39: number analyzed (Participants) | 24 | 39
  Lymphocytes:Week 12; n=24, 39 | 0.098 (0.3657) | 0.044 (0.3546)
  Lymphocytes:Week 14; n=23, 39: number analyzed (Participants) | 23 | 39
  Lymphocytes:Week 14; n=23, 39 | 0.009 (0.3590) | 0.119 (0.4346)
  Lymphocytes:Week 16; n=23, 39: number analyzed (Participants) | 23 | 39
  Lymphocytes:Week 16; n=23, 39 | 0.02 (0.3825) | 0.075 (0.4397)
  Lymphocytes:Week 28; n=65, 60: number analyzed (Participants) | 65 | 60
  Lymphocytes:Week 28; n=65, 60 | 0.065 (0.4601) | 0.162 (0.4794)
  Neutrophils: Week 1; n=77, 74: number analyzed (Participants) | 77 | 74
  Neutrophils: Week 1; n=77, 74 | 0.079 (1.4665) | 0.092 (1.1019)
  Neutrophils:Week 2; n=68, 72: number analyzed (Participants) | 68 | 72
  Neutrophils:Week 2; n=68, 72 | 0.023 (1.0414) | 0.035 (0.8299)
  Neutrophils:Week 4; n=48, 57: number analyzed (Participants) | 48 | 57
  Neutrophils:Week 4; n=48, 57 | 0.187 (1.2738) | 0.217 (1.2788)
  Neutrophils:Week 6; n=43, 54: number analyzed (Participants) | 43 | 54
  Neutrophils:Week 6; n=43, 54 | 0.203 (1.3952) | -0.126 (0.8524)
  Neutrophils:Week 8; n=33, 46: number analyzed (Participants) | 33 | 46
  Neutrophils:Week 8; n=33, 46 | -0.080 (0.9654) | 0.331 (2.0776)
  Neutrophils:Week 10; n=32, 44: number analyzed (Participants) | 32 | 44
  Neutrophils:Week 10; n=32, 44 | -0.192 (0.9739) | 0.041 (0.9173)
  Neutrophils:Week 12; n=24, 39: number analyzed (Participants) | 24 | 39
  Neutrophils:Week 12; n=24, 39 | -0.013 (1.2306) | 0.158 (0.8630)
  Neutrophils:Week 14; n=23, 39: number analyzed (Participants) | 23 | 39
  Neutrophils:Week 14; n=23, 39 | -0.263 (1.3117) | 0.073 (0.9305)
  Neutrophils:Week 16; n=23, 39: number analyzed (Participants) | 23 | 39
  Neutrophils:Week 16; n=23, 39 | -0.448 (1.1201) | 0.142 (1.2595)
  Neutrophils:Week 28; n=65, 60: number analyzed (Participants) | 65 | 60
  Neutrophils:Week 28; n=65, 60 | -0.201 (1.5148) | -0.045 (1.1145)
  Monocytes: Week 1; n=77, 74: number analyzed (Participants) | 77 | 74
  Monocytes: Week 1; n=77, 74 | 0.026 (0.1595) | 0.015 (0.1209)
  Monocytes:Week 2; n=68, 72: number analyzed (Participants) | 68 | 72
  Monocytes:Week 2; n=68, 72 | 0.020 (0.1226) | 0.022 (0.0965)
  Monocytes:Week 4; n=48, 57: number analyzed (Participants) | 48 | 57
  Monocytes:Week 4; n=48, 57 | 0.051 (0.1869) | 0.027 (0.1014)
  Monocytes:Week 6; n=43, 54: number analyzed (Participants) | 43 | 54
  Monocytes:Week 6; n=43, 54 | 0.050 (0.1353) | 0.038 (0.1083)
  Monocytes:Week 8; n=33, 46: number analyzed (Participants) | 33 | 46
  Monocytes:Week 8; n=33, 46 | 0.045 (0.1152) | 0.023 (0.1038)
  Monocytes:Week 10; n=32, 44: number analyzed (Participants) | 32 | 44
  Monocytes:Week 10; n=32, 44 | 0.090 (0.1463) | 0.038 (0.100)
  Monocytes:Week 12; n=24, 39: number analyzed (Participants) | 24 | 39
  Monocytes:Week 12; n=24, 39 | 0.073 (0.1362) | 0.025 (0.0948)
  Monocytes:Week 14; n=23, 39: number analyzed (Participants) | 23 | 39
  Monocytes:Week 14; n=23, 39 | 0.059 (0.1301) | 0.082 (0.103)
  Monocytes:Week 16; n=23, 39: number analyzed (Participants) | 23 | 39
  Monocytes:Week 16; n=23, 39 | 0.040 (0.1087) | 0.053 (0.1075)
  Monocytes:Week 28; n=65, 60: number analyzed (Participants) | 65 | 60
  Monocytes:Week 28; n=65, 60 | 0.041 (0.1431) | 0.066 (0.1218)
  Platelets: Week 1; n=78, 74 | 1.5 (31.89) | 8.7 (44.52)
  Platelets:Week 2; n=71, 74: number analyzed (Participants) | 71 | 74
  Platelets:Week 2; n=71, 74 | 7.6 (35.72) | 9.8 (44.42)
  Platelets:Week 4; n=49, 57: number analyzed (Participants) | 49 | 57
  Platelets:Week 4; n=49, 57 | 4.0 (27.64) | 5.3 (33.05)
  Platelets:Week 6; n=44, 56: number analyzed (Participants) | 44 | 56
  Platelets:Week 6; n=44, 56 | 18.2 (46.02) | 3.9 (35.62)
  Platelets:Week 8; n=34, 47: number analyzed (Participants) | 34 | 47
  Platelets:Week 8; n=34, 47 | 8.6 (38.79) | -1.1 (30.31)
  Platelets:Week 10; n=34, 45: number analyzed (Participants) | 34 | 45
  Platelets:Week 10; n=34, 45 | 10.9 (45.93) | 4.7 (30.88)
  Platelets:Week 12; n=24, 39: number analyzed (Participants) | 24 | 39
  Platelets:Week 12; n=24, 39 | 3.6 (46.24) | 6.6 (27.79)
  Platelets:Week 14; n=24, 39: number analyzed (Participants) | 24 | 39
  Platelets:Week 14; n=24, 39 | -6.4 (45.37) | 5.5 (32.66)
  Platelets:Week 16; n=24, 38: number analyzed (Participants) | 24 | 38
  Platelets:Week 16; n=24, 38 | -0.5 (37.57) | 6.3 (40.13)
  Platelets:Week 28; n=64, 62: number analyzed (Participants) | 64 | 62
  Platelets:Week 28; n=64, 62 | -3.5 (35.52) | 3.0 (52.16)

40. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocyte Mean Corpuscular Volume
Description: Blood samples were collected for the analysis of erythrocyte mean corpuscular volume at indicated time points.Baseline is defined as the most recent recorded value before dosing on Day 1. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline and Weeks1, 2, 4, 6, 8, 10, 12, 14, 16 and 28
Population: Safety Population. Only those participants with data available at indicated time points were analyzed . Participants with data available at specified time points were represented by n=x in the category titles.
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 78 | 74
Femtoliters
  Week 1: n=78,74 | 0.3 (1.59) | -0.1 (1.46)
  Week 2: n=71, 74: number analyzed (Participants) | 71 | 74
  Week 2: n=71, 74 | 0.2 (1.44) | -0.2 (1.62)
  Week 4: n=49, 57: number analyzed (Participants) | 49 | 57
  Week 4: n=49, 57 | -0.4 (1.62) | -0.6 (1.98)
  Week 6: n=44, 56: number analyzed (Participants) | 44 | 56
  Week 6: n=44, 56 | -0.3 (1.29) | -0.4 (2.33)
  Week 8: n=34, 47: number analyzed (Participants) | 34 | 47
  Week 8: n=34, 47 | -0.9 (1.37) | -0.6 (2.13)
  Week 10: n=34, 45: number analyzed (Participants) | 34 | 45
  Week 10: n=34, 45 | -1.1 (1.82) | -0.9 (2.52)
  Week 12: n=24, 39: number analyzed (Participants) | 24 | 39
  Week 12: n=24, 39 | -0.7 (1.46) | -1.3 (2.61)
  Week 14: n=24, 39: number analyzed (Participants) | 24 | 39
  Week 14: n=24, 39 | -0.7 (1.63) | -1.5 (2.46)
  Week 16: n=24, 39: number analyzed (Participants) | 24 | 39
  Week 16: n=24, 39 | -0.6 (1.58) | -2.3 (2.67)
  Week 28: n=65, 63: number analyzed (Participants) | 65 | 63
  Week 28: n=65, 63 | -1.6 (2.76) | -2.9 (5.20)

41. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes
Description: Blood samples were collected for the analysis of erythrocytes at indicated time points. Baseline is defined as the most recent recorded value before dosing on Day 1. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline and Weeks 1, 2, 4, 6, 8, 10, 12, 14, 16 and 28
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 78 | 74
10^12 cells per liter
  Week 1: n=78,74 | -0.01 (0.220) | -0.03 (0.232)
  Week 2: n=71, 74: number analyzed (Participants) | 71 | 74
  Week 2: n=71, 74 | 0.01 (0.232) | 0.01 (0.200)
  Week 4: n=49, 57: number analyzed (Participants) | 49 | 57
  Week 4: n=49, 57 | 0.05 (0.298) | -0.01 (0.169)
  Week 6: n=44, 56: number analyzed (Participants) | 44 | 56
  Week 6: n=44, 56 | 0.05 (0.181) | -0.04 (0.170)
  Week 8: n=34, 47: number analyzed (Participants) | 34 | 47
  Week 8: n=34, 47 | 0.02 (0.210) | 0.02 (0.234)
  Week 10: n=34, 45: number analyzed (Participants) | 34 | 45
  Week 10: n=34, 45 | 0.00 (0.228) | -0.02 (0.201)
  Week 12: n=24, 39: number analyzed (Participants) | 24 | 39
  Week 12: n=24, 39 | 0.06 (0.226) | -0.03 (0.297)
  Week 14: n=24, 39: number analyzed (Participants) | 24 | 39
  Week 14: n=24, 39 | 0.03 (0.206) | 0.04 (0.253)
  Week 16: n=24, 39: number analyzed (Participants) | 24 | 39
  Week 16: n=24, 39 | 0.00 (0.184) | 0.03 (0.236)
  Week 28: n=65, 63: number analyzed (Participants) | 65 | 63
  Week 28: n=65, 63 | 0.09 (0.260) | 0.09 (0.381)

42. Secondary Outcome: Change From Baseline in Hematology Parameter: Hemoglobin
Description: Blood samples were collected for the analysis of hemoglobin level at indicated time points. Baseline is defined as the most recent recorded value before dosing on Day 1. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline and Weeks1, 2, 4, 6, 8, 10, 12, 14, 16 and 28
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 78 | 74
Grams per liter
  Week 1: n=78,74 | 0.5 (7.08) | -0.7 (6.30)
  Week 2: n=71, 74: number analyzed (Participants) | 71 | 74
  Week 2: n=71, 74 | 0.5 (7.01) | 0.0 (5.64)
  Week 4: n=49, 57: number analyzed (Participants) | 49 | 57
  Week 4: n=49, 57 | 1.6 (8.84) | -0.4 (5.16)
  Week 6: n=44, 56: number analyzed (Participants) | 44 | 56
  Week 6: n=44, 56 | 1.5 (4.60) | -1.2 (5.17)
  Week 8: n=34, 47: number analyzed (Participants) | 34 | 47
  Week 8: n=34, 47 | 0.5 (6.16) | -0.1 (6.72)
  Week 10: n=34, 45: number analyzed (Participants) | 34 | 45
  Week 10: n=34, 45 | -0.4 (5.71) | -0.8 (5.28)
  Week 12: n=24, 39: number analyzed (Participants) | 24 | 39
  Week 12: n=24, 39 | 1.0 (6.50) | -1.8 (10.05)
  Week 14: n=24, 39: number analyzed (Participants) | 24 | 39
  Week 14: n=24, 39 | -0.6 (6.08) | -0.3 (6.35)
  Week 16: n=24, 39: number analyzed (Participants) | 24 | 39
  Week 16: n=24, 39 | -0.5 (5.44) | 0.0 (6.14)
  Week 28: n=65, 63: number analyzed (Participants) | 65 | 63
  Week 28: n=65, 63 | 1.0 (8.20) | -0.7 (10.24)

43. Secondary Outcome: Change From Baseline in Hematology Parameter: Hematocrit Level
Description: Blood samples were collected for the analysis of hematocrit at indicated time points. Baseline is defined as the most recent recorded value before dosing on Day 1. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline and Weeks 1, 2, 4, 6, 8, 10, 12, 14, 16 and 28
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 78 | 74
Proportion of red blood cells in blood
  Week 1: n=78,74 | 0.0007 (0.02255) | -0.0025 (0.02114)
  Week 2: n=71, 74: number analyzed (Participants) | 71 | 74
  Week 2: n=71, 74 | 0.0024 (0.02213) | -0.0046 (0.04223)
  Week 4: n=49, 57: number analyzed (Participants) | 49 | 57
  Week 4: n=49, 57 | 0.0038 (0.02957) | -0.0033 (0.01665)
  Week 6: n=44, 56: number analyzed (Participants) | 44 | 56
  Week 6: n=44, 56 | 0.0024 (0.01557) | -0.0050 (0.02060)
  Week 8: n=34, 47: number analyzed (Participants) | 34 | 47
  Week 8: n=34, 47 | -0.0019 (0.01645) | -0.0015 (0.02212)
  Week 10: n=34, 45: number analyzed (Participants) | 34 | 45
  Week 10: n=34, 45 | -0.0050 (0.01897) | -0.0061 (0.02175)
  Week 12: n=24, 39: number analyzed (Participants) | 24 | 39
  Week 12: n=24, 39 | 0.0009 (0.01740) | -0.0088 (0.03342)
  Week 14: n=24, 39: number analyzed (Participants) | 24 | 39
  Week 14: n=24, 39 | -0.0018 (0.01699) | -0.0038 (0.02277)
  Week 16: n=24, 39: number analyzed (Participants) | 24 | 39
  Week 16: n=24, 39 | -0.0042 (0.01474) | -0.0071 (0.02232)
  Week 28: n=65, 63: number analyzed (Participants) | 65 | 63
  Week 28: n=65, 63 | 0.0016 (0.02283) | -0.0041 (0.03153)

44. Secondary Outcome: Change From Baseline in Hematology Parameter: Mean Corpuscular Hemoglobin
Description: Blood samples were collected for the analysis of mean corpuscular hemoglobin at indicated time points. Baseline is defined as the most recent recorded value before dosing on Day 1. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline and Weeks 1, 2, 4, 6, 8, 10, 12, 14, 16 and 28
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Picogram
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 78 | 74
Picogram
  Week 1: n=78,74 | 0.17 (0.725) | 0.01 (0.453)
  Week 2: n=71, 74: number analyzed (Participants) | 71 | 74
  Week 2: n=71, 74 | 0.01 (0.430) | -0.07 (0.471)
  Week 4: n=49, 57: number analyzed (Participants) | 49 | 57
  Week 4: n=49, 57 | 0.01 (0.461) | -0.04 (0.432)
  Week 6: n=44, 56: number analyzed (Participants) | 44 | 56
  Week 6: n=44, 56 | 0.06 (0.416) | 0.00 (0.551)
  Week 8: n=34, 47: number analyzed (Participants) | 34 | 47
  Week 8: n=34, 47 | 0.02 (0.660) | -0.11 (0.567)
  Week 10: n=34, 45: number analyzed (Participants) | 34 | 45
  Week 10: n=34, 45 | -0.06 (0.590) | -0.01 (0.863)
  Week 12: n=24, 39: number analyzed (Participants) | 24 | 39
  Week 12: n=24, 39 | -0.07 (0.543) | -0.12 (0.776)
  Week 14: n=24, 39: number analyzed (Participants) | 24 | 39
  Week 14: n=24, 39 | -0.23 (0.421) | -0.29 (0.785)
  Week 16: n=24, 39: number analyzed (Participants) | 24 | 39
  Week 16: n=24, 39 | -0.05 (0.475) | -0.26 (0.839)
  Week 28: n=65, 63: number analyzed (Participants) | 65 | 63
  Week 28: n=65, 63 | -0.40 (0.649) | -0.78 (1.773)

45. Secondary Outcome: Change From Baseline in Hematology Parameter: Mean Corpuscular Hemoglobin Concentration
Description: Blood samples were collected for the analysis of mean corpuscular hemoglobin concentration at indicated time points.Baseline is defined as the most recent recorded value before dosing on Day 1. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline and Weeks 1, 2, 4, 6, 8, 10, 12, 14, 16 and 28
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 78 | 74
Grams per liter
  Week 1: n=78,74 | 0.8 (8.29) | 0.5 (6.65)
  Week 2: n=71, 74: number analyzed (Participants) | 71 | 74
  Week 2: n=71, 74 | -0.6 (6.04) | 0.2 (7.09)
  Week 4: n=49, 57: number analyzed (Participants) | 49 | 57
  Week 4: n=49, 57 | 1.2 (7.01) | 1.5 (7.32)
  Week 6: n=44, 56: number analyzed (Participants) | 44 | 56
  Week 6: n=44, 56 | 1.9 (5.33) | 1.3 (9.33)
  Week 8: n=34, 47: number analyzed (Participants) | 34 | 47
  Week 8: n=34, 47 | 3.0 (7.65) | 1.1 (7.56)
  Week 10: n=34, 45: number analyzed (Participants) | 34 | 45
  Week 10: n=34, 45 | 3.3 (6.68) | 3.4 (10.17)
  Week 12: n=24, 39: number analyzed (Participants) | 24 | 39
  Week 12: n=24, 39 | 2.3 (6.29) | 3.2 (10.32)
  Week 14: n=24, 39: number analyzed (Participants) | 24 | 39
  Week 14: n=24, 39 | 0.4 (6.47) | 2.4 (8.97)
  Week 16: n=24, 39: number analyzed (Participants) | 24 | 39
  Week 16: n=24, 39 | 2.1 (7.01) | 5.7 (9.60)
  Week 28: n=65, 63: number analyzed (Participants) | 65 | 63
  Week 28: n=65, 63 | 1.2 (8.36) | 1.5 (8.78)

46. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes Distribution Width (%)
Description: Blood samples were collected for the analysis of Erythrocytes Distribution Width (%) at indicated time points. Baseline is defined as the most recent recorded value before dosing on Day 1. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline and Weeks1, 2, 4, 6, 8, 10, 12, 14, 16 and 28
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Percentage (%) of Erythrocytes
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 78 | 74
Percentage (%) of Erythrocytes
  Week 1: n=78,74 | -0.06 (0.747) | -0.08 (0.604)
  Week 2: n=71, 74: number analyzed (Participants) | 71 | 74
  Week 2: n=71, 74 | -0.02 (0.478) | -0.20 (0.652)
  Week 4: n=49, 57: number analyzed (Participants) | 49 | 57
  Week 4: n=49, 57 | -0.22 (0.555) | -0.33 (0.844)
  Week 6: n=44, 56: number analyzed (Participants) | 44 | 56
  Week 6: n=44, 56 | -0.33 (0.545) | -0.37 (0.861)
  Week 8: n=34, 47: number analyzed (Participants) | 34 | 47
  Week 8: n=34, 47 | -0.40 (0.669) | -0.29 (0.960)
  Week 10: n=34, 45: number analyzed (Participants) | 34 | 45
  Week 10: n=34, 45 | -0.35 (0.791) | -0.38 (1.049)
  Week 12: n=24, 39: number analyzed (Participants) | 24 | 39
  Week 12: n=24, 39 | -0.27 (0.717) | -0.34 (0.916)
  Week 14: n=24, 39: number analyzed (Participants) | 24 | 39
  Week 14: n=24, 39 | -0.28 (0.873) | -0.38 (0.897)
  Week 16: n=24, 39: number analyzed (Participants) | 24 | 39
  Week 16: n=24, 39 | -0.25 (0.727) | -0.41 (0.995)
  Week 28: n=65, 63: number analyzed (Participants) | 65 | 63
  Week 28: n=65, 63 | -0.09 (1.028) | -0.01 (1.202)

47. Secondary Outcome: Change From Baseline in Cardiac Marker: N-Terminal ProB-type Natriuretic Peptide
Description: Blood samples were collected for the analysis of N-Terminal ProB-type Natriuretic Peptide at indicated time points.Baseline is defined as the most recent recorded value before dosing on Day 1. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline and Weeks 1, 2, 4, 6, 8, 10, 12, 14, 16 and 28
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Nanograms per liter
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 79 | 75
Nanograms per liter
  Week 1: n=79,75 | -14.8442 (61.92992) | 8.4023 (54.37938)
  Week 2: n=73,75: number analyzed (Participants) | 73 | 75
  Week 2: n=73,75 | -10.8134 (71.40009) | -2.5196 (42.06499)
  Week 4: n=49, 59: number analyzed (Participants) | 49 | 59
  Week 4: n=49, 59 | -17.9849 (68.85651) | -4.5560 (44.12297)
  Week 6: n=45, 57: number analyzed (Participants) | 45 | 57
  Week 6: n=45, 57 | -5.0620 (53.06025) | 3.6194 (53.96329)
  Week 8: n=34, 47: number analyzed (Participants) | 34 | 47
  Week 8: n=34, 47 | -8.6398 (49.58134) | 9.6509 (66.34546)
  Week 10: n=34, 46: number analyzed (Participants) | 34 | 46
  Week 10: n=34, 46 | -12.7377 (80.51666) | 14.9119 (58.17102)
  Week 12: n=24, 38: number analyzed (Participants) | 24 | 38
  Week 12: n=24, 38 | -13.6951 (53.70314) | 8.8531 (58.15689)
  Week 14: n=24, 39: number analyzed (Participants) | 24 | 39
  Week 14: n=24, 39 | -4.8082 (57.47926) | 20.0149 (74.94234)
  Week 16: n=24, 39: number analyzed (Participants) | 24 | 39
  Week 16: n=24, 39 | -19.4899 (58.89689) | 4.7760 (60.56438)
  Week 28: n=65, 65: number analyzed (Participants) | 65 | 65
  Week 28: n=65, 65 | -6.1970 (62.26132) | 0.9810 (64.44446)

48. Secondary Outcome: Change From Baseline in Cardiac Marker: Cardiac Troponin I
Description: Blood samples were collected for the analysis of Troponin I at indicated time points.Baseline is defined as the most recent recorded value before dosing on Day 1. Change from Baseline was calculated by subtracting Baseline value from the specified time point value.
Time Frame: Baseline and Weeks 1, 2, 4, 6, 8, 10, 12, 14, 16 and 28
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: Micrograms per liter
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 78 | 74
Micrograms per liter
  Week 1: n=78,74 | 0.000 (0.0000) | 0.000 (0.0023)
  Week 2: n=73, 73: number analyzed (Participants) | 73 | 73
  Week 2: n=73, 73 | 0.000 (0.0016) | 0.000 (0.0023)
  Week 4: n=49, 58: number analyzed (Participants) | 49 | 58
  Week 4: n=49, 58 | 0.001 (0.0059) | 0.000 (0.0000)
  Week 6: n=45, 57: number analyzed (Participants) | 45 | 57
  Week 6: n=45, 57 | 0.000 (0.0021) | 0.000 (0.0000)
  Week 8: n=34, 46: number analyzed (Participants) | 34 | 46
  Week 8: n=34, 46 | 0.000 (0.0017) | 0.000 (0.0000)
  Week 10: n=34, 38: number analyzed (Participants) | 34 | 38
  Week 10: n=34, 38 | 0.006 (0.0344) | 0.000 (0.0000)
  Week 12: n=24, 39: number analyzed (Participants) | 24 | 39
  Week 12: n=24, 39 | 0.000 (0.0000) | 0.000 (0.0000)
  Week 14: n=24, 39: number analyzed (Participants) | 24 | 39
  Week 14: n=24, 39 | 0.000 (0.0000) | 0.000 (0.0016)
  Week 16: n=24, 39: number analyzed (Participants) | 24 | 39
  Week 16: n=24, 39 | 0.000 (0.0000) | 0.000 (0.0000)
  Week 28: n=63, 63: number analyzed (Participants) | 63 | 63
  Week 28: n=63, 63 | 0.000 (0.0013) | -0.001 (0.0050)

49. Secondary Outcome: Number of Participants With Incidence and Titres of Anti- GSK3772847 Antibodies
Description: Blood samples were collected at given time points and the presence of anti-GSK3772847 antibodies were assessed using a a tiered approach including a screening assay, a confirmation assay and calculation of titer. Data for participants who showed positive results for confirmation assay has been presented
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24 and 28
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 74 | 75
Participants
  Week2; n=73, 74: number analyzed (Participants) | 73 | 74
  Week2; n=73, 74 | 0 | 0
  Week4; n=49, 59: number analyzed (Participants) | 49 | 59
  Week4; n=49, 59 | 0 | 0
  Week8; n=34, 47: number analyzed (Participants) | 34 | 47
  Week8; n=34, 47 | 0 | 0
  Week12; n=24, 39: number analyzed (Participants) | 24 | 39
  Week12; n=24, 39 | 0 | 0
  Week16; n=23, 39: number analyzed (Participants) | 23 | 39
  Week16; n=23, 39 | 0 | 0
  Week20; n=73, 75: number analyzed (Participants) | 73 | 75
  Week20; n=73, 75 | 1 | 0
  Week24; n=74, 75 | 0 | 0
  Week28; n=74, 74: number analyzed (Participants) | 74 | 74
  Week28; n=74, 74 | 0 | 0

50. Secondary Outcome: Serum Concentrations of GSK3772847
Description: Blood samples were collected at given time points to evaluate pharmacokinetics (PK) of GSK3772847 in participants with moderately severe asthma.
Time Frame: Weeks 2, 4 (Pre-dose), 8 (Pre-dose), 12 (Pre-dose and Post-dose), 16, 20, 24 and 28
Population: PK Population consists of all randomized participants who received at least one dose of study medication, and for whom at least one pharmacokinetic sample was obtained, analyzed and was measurable. Participants with data available at specified time points were represented by n=x in the category titles.
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter
Arm/Group | GSK3772847
Number analyzed (Participants) | 75
Micrograms per milliliter
  Week2; n=75 | 78.40 (30.934)
  Week4; Pre-dose;n=59: number analyzed (Participants) | 59
  Week4; Pre-dose;n=59 | 44.42 (21.774)
  Week8; Pre-dose; n= 47: number analyzed (Participants) | 47
  Week8; Pre-dose; n= 47 | 61.44 (30.978)
  Week12; Pre-dose; n=39: number analyzed (Participants) | 39
  Week12; Pre-dose; n=39 | 63.42 (34.420)
  Week12; Post-dose; n=39: number analyzed (Participants) | 39
  Week12; Post-dose; n=39 | 224.21 (151.780)
  Week16; n=38: number analyzed (Participants) | 38
  Week16; n=38 | 63.03 (36.328)
  Week20; n=75 | 25.75 (19.074)
  Week24; n=75 | 12.91 (16.061)
  Week28; n=75 | 6.14 (16.005)

51. Secondary Outcome: Percent Change From Baseline in Free Soluble Suppressor of Tumorigenicity 2 (ST2) Concentration
Description: Blood samples were collected at given time points to measure free soluble ST2 concentration. Baseline is defined as the latest available assessment prior to first dose (Day 1). Analysis was performed using mixed model repeated measures. Percent change from Baseline is calculated as ratio to Baseline minus 1 and multiplied by 100.
Time Frame: Baseline and Week 4 (Pre-dose), Week 8 (Pre-dose), Week 12 (Pre-dose) and Week 16
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 78 | 78
Percent change
  Week4; Pre-dose; n=48, 56: number analyzed (Participants) | 48 | 56
  Week4; Pre-dose; n=48, 56 | -5.6 [-20.8 to 12.4] | -93.8 [-94.7 to -92.7]
  Week8; Pre-dose; n=33, 45: number analyzed (Participants) | 33 | 45
  Week8; Pre-dose; n=33, 45 | -8.5 [-26.9 to 14.5] | -93.5 [-94.7 to -92.0]
  Week12; Pre-dose; n=23, 37: number analyzed (Participants) | 23 | 37
  Week12; Pre-dose; n=23, 37 | 10.5 [-17.4 to 47.7] | -92.5 [-94.2 to -90.4]
  Week16; n=16, 26: number analyzed (Participants) | 16 | 26
  Week16; n=16, 26 | 19.8 [-8.8 to 57.3] | -92.0 [-93.7 to -89.9]
Statistical Analysis 1: Comparison: Placebo vs GSK3772847; Test type: Other; p < 0.001, mixed model repeated measures analysis — Week 4; Percent change = -93.4, 95% CI 2-sided [-94.9 to -91.7]
Statistical Analysis 2: Comparison: Placebo vs GSK3772847; Test type: Other; p < 0.001, mixed model repeated measures analysis — Week 8; Percent change = -92.9, 95% CI 2-sided [-94.8 to -90.3]
Statistical Analysis 3: Comparison: Placebo vs GSK3772847; Test type: Other; p < 0.001, mixed model repeated measures analysis — Week 12; Percent change = -93.2, 95% CI 2-sided [-95.4 to -90.0]
Statistical Analysis 4: Comparison: Placebo vs GSK3772847; Test type: Other; p < 0.001, mixed model repeated measures analysis — Week 16; Percent change = -93.3, 95% CI 2-sided [-95.3 to -90.4]

52. Secondary Outcome: Percent Change From Baseline in Total Soluble ST2 Concentration
Description: Blood samples were collected at given time points to measure total soluble ST2 concentration. Baseline is defined as the latest available assessment prior to first dose (Day 1). Analysis was performed using mixed model repeated measures. Percent change from Baseline is calculated as ratio to Baseline minus 1 and multiplied by 100.
Time Frame: Baseline and Week 4 (Pre-dose), Week 8 (Pre-dose), Week 12 (Pre-dose) and Week 16
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo | GSK3772847
Number analyzed (Participants) | 48 | 56
Percent change
  Week4; Pre-dose; n=48, 56 | 16.3 [-0.6 to 36.0] | 2691.1 [2314.4 to 3126.6]
  Week8; Pre-dose; n=33, 45: number analyzed (Participants) | 33 | 45
  Week8; Pre-dose; n=33, 45 | -6.9 [-22.7 to 12.0] | 2326.9 [1951.7 to 2770.7]
  Week12; Pre-dose; n=23, 37: number analyzed (Participants) | 23 | 37
  Week12; Pre-dose; n=23, 37 | -13.4 [-33.4 to 12.6] | 1858.0 [1461.4 to 2355.2]
  Week16; n=16, 26: number analyzed (Participants) | 16 | 26
  Week16; n=16, 26 | -12.0 [-28.5 to 8.3] | 2330.8 [1933.0 to 2806.4]
Statistical Analysis 1: Comparison: Placebo vs GSK3772847; Test type: Other; p < 0.001, mixed model repeated measures analysis — Week 4; Percent change = 2300.4, 95% CI 2-sided [1833.9 to 2879.3]
Statistical Analysis 2: Comparison: Placebo vs GSK3772847; Test type: Other; p < 0.001, mixed model repeated measures analysis — Week 8; Percent change = 2507.7, 95% CI 2-sided [1924.2 to 3259.4]
Statistical Analysis 3: Comparison: Placebo vs GSK3772847; Test type: Other; p < 0.001, mixed model repeated measures analysis — Week 12; Percent change = 2162.2, 95% CI 2-sided [1489.1 to 3120.3]
Statistical Analysis 4: Comparison: Placebo vs GSK3772847; Test type: Other; p < 0.001, mixed model repeated measures analysis — Week 16; Percent change = 2663.0, 95% CI 2-sided [1994.6 to 3544.8]

ADVERSE EVENTS:
Time Frame: SAEs and non-SAEs were collected for 16 weeks.
Description: SAEs and non-SAEs were reported for Safety Population. The non-SAEs were reported using a frequency threshold of >=3%.
Arm/Group | Placebo | GSK3772847
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/83
Serious Adverse Events (participants affected / at risk) | 1/82 | 2/83
Other Adverse Events (participants affected / at risk) | 20/82 | 19/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=82) | GSK3772847 (N=83)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=82) | GSK3772847 (N=83)
Nasopharyngitis (Infections and infestations) | 4 (5) | 4 (6)
Influenza (Infections and infestations) | 4 (4) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 4 (5)
Headache (Nervous system disorders) | 9 (15) | 9 (17)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (5)
Ventricular tachycardia (Cardiac disorders) | 3 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-09-13): https://cdn.clinicaltrials.gov/large-docs/43/NCT03207243/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-27): https://cdn.clinicaltrials.gov/large-docs/43/NCT03207243/SAP_001.pdf